

Title: A Single-Arm, Multicenter, Phase 2 Study of Brigatinib in Japanese Patients With ALK-Positive Non-Small Cell Lung Cancer (NSCLC)

NCT Number: NCT03410108

Statistical analysis plan Approve Date: 13-Jul-2020

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).



# STATISTICAL ANALYSIS PLAN

STUDY NUMBER: Brigatinib-2001

the applicable remisorilise lients A Single-Arm, Multicenter, Phase 2 Study of Brigatinib in Japanese Patients With ALK-Positive Non-Small Cell Lung Cancer (NSCLC)

# PHASE 2

Version: Amendment 6

Date: 13 Jul 2021

Prepared by:

Based on:

Protocol Version: Amendment 4

Protocol Date: 22 Jul 2020

Properly of Takeda: For non-commercial use only and subject to the applicable Terms of use

| 2.0 | TABLE | E OF CONTENTS | |
|---|---|---|---|
| 1.0 | TITLE | PAGE | 1 |
| 1. | 1 App | roval Signatures | 2 |
| 2.0 | TABLE | OF CONTENTS | <u>3</u> |
| 3.0 | LIST O | F ABBREVIATIONS | 6 |
| 4.0 | OBJEC | TIVES | 9 |
| 4. | 1 Prin | nary Objectives | 9 |
| 4. | 2 Seco | ondary Objectives | 9 |
| 4. | 3 Safe | F ABBREVIATIONS TIVES nary Objectives ondary Objectives ety Objectives | 9 |
| 4. | 4 | | |
| 4. | 5 Stud | ly Design | 9 |
| 5.0 | ANALY | YSIS ENDPOINTS | .12 |
| 5. | 1 Prin | dy Design YSIS ENDPOINTS nary Endpoint ondary Endpoints ety Endpoints | .12 |
| 5 | 2 Seco | ondary Endpoints | .12 |
| 5 | 3 Safe | ety Endpoints | .13 |
| 5. | 4 | | 13 |
| 6.0 | | MINATION OF SAMPLE SIZE | |
| 7.0 | METHO | ODS OF ANALYSIS AND PRESENTATION | .15 |
| 7. | 1 Gen | eral Principles | .15 |
| | 7.1.1 | Study Definitions. | .15 |
| | 7.1.2 | Definition of Study Days | .19 |
| | 7.1.3 | Definition of Study Visit Windows | .19 |
| | 7.1.4 | Methods for Handling Missing Data and Specific Data | |
| 7. | 2 Ana | lysis Sets | .21 |
| 7. | _ | position of Subjects | |
| | 7.3.1 | Study Information | .23 |
| | 7.3.2 | Screen Failures | .23 |
| | 73.3 | Subject Eligibility | |
| . < | ٥ <sup>7</sup> .3.4 | Number of Subjects Who Entered the Treatment Period by Site | |
| Ŏ, | 7.3.5 | Disposition of Subjects | |
| } | 7.3.6 | Protocol Deviations | .25 |
| | 7.3.7 | Analysis Sets | |
| 7. | | nographic and Other Baseline Characteristics | |
| 7. | | dical History and Concurrent Medical Conditions | |
| 7. | 6 Med | lication History and Concomitant Medications | .30 |

| Brigatinib-2001<br>Statistical Analy | vsis Plan Amendment 6 | Page 4 of 83<br>13 Jul 2021 |
|---|---|---|
| 7.7 Stu | dy Drug Exposure and Compliance | 30 |
| | icacy Analysis | 31 |
| 7.8.1 | Primary Efficacy Endpoint(s) | 31 |
| 7.8.2 | Primary Efficacy Endpoint(s) | |
| 7.8.3 | Additional Efficacy Endpoint(s) armacokinetic/Pharmacodynamic Analysis Pharmacokinetic Analysis Pharmacodynamic Analysis ner Outcomes Sety Analysis | 36 |
| 7.9 Pha | armacokinetic/Pharmacodynamic Analysis | 38 |
| 7.9.1 | Pharmacokinetic Analysis | 38 |
| 7.9.2 | Pharmacodynamic Analysis | 39 |
| 7.10 Otl | ner Outcomes | 40 |
| 7.11 Sat | ety Analysis | 40 |
| 7.11.1 | Adverse Events | 40 |
| 7.11.2 | Clinical Laboratory Evaluations | 56 |
| 7.11.3 | Vital Signs | 57 |
| 7.11.4 | 12-Lead ECGs | 58 |
| 7.11.5 | Other Observations Related to Safety | 59 |
| 7.12 Int | Adverse Events Clinical Laboratory Evaluations Vital Signs 12-Lead ECGs Other Observations Related to Safety erim Analysis Analysis plan at the Interim Analysis | 59 |
| 7.12.1 | Analysis plan at the Interim Analysis | 60 |
| 7.12.2 | Analysis plan in safety lead-in part | 60 |
| 7.13 Pla | nned Analysis for the Refractory Patients and one for TKI-naïve Patient | s61 |
| 7.13.1 | Planned Analysis for the Refractory Patients | 61 |
| 7.13.2 | Planned Analysis for TKI-naïve Patients | |
| 7.13.3 | Planned Final Analysis | 61 |
| 7.14 Ch | anges in the Statistical Analysis Plan | 61 |
| 8.0 REFEI | RENCES | 62 |
| | 70, | |
| LIST OF IN- | TEXT TABLES | |
| * | The Scheme of Progression and Censoring for PFS | 16 |
| Table 7.8 | Minimum Number of Confirmed ORR at the Primary Analysis | |
| 13/ | , | |
| EIST OF IN- | TEXT FIGURES | |
| Figure 4.a | Overview of Study Design | 11 |

#### 3.0 LIST OF ABBREVIATIONS

ΑE adverse event

ALK anaplastic lymphoma kinase

A JSE ONLY and Subject to the applicable Terms of Use ALP alkaline phosphatase ALT alanine aminotransferase **ANC** absolute neutrophil count AST aspartate aminotransferase

**AUC** area under the plasma concentration-time curve

BID twice daily

**BUN** blood urea nitrogen CL/F oral clearance

 $C_{\text{max}}$ maximum observed plasma concentration

**CNS** central nervous system **CPK** creatine phosphokinase CR complete response

**CRO** contract research organization

**CSR** clinical study report CTcomputed tomography ctDNA circulating tumor DNA

CxDx Cycle x Day x **CYP** cytochrome P450 **DCR** disease control rate drug-drug interaction DDI

Dohmen Life Science Services **DLSS** 

DLT dose-limiting toxicity duration of response DOR electrocardiogram **ECG** 

**ECOG** Eastern Cooperative Oncology Group

eCRF electronic case report form **EGFR** epidermal growth factor receptor **EOPE** early onset pulmonary event

**EORTC** European Organisation for Research and Treatment of Cancer

end of treatment

EQ-5D-5L the 5-level version of the EuroQol 5-dimensional questionnaire

European Union full analysis set

Food and Drug Administration **FFPE** formalin-fixed, paraffin-embedded **FISH** fluorescence in situ hybridization

**GCP** Good Clinical Practice G-CSF

**GM-CSF** 

HbA1c

**HBcAb** HBsAb **HBsAg** 

**HBV HCV** 

**HCVAb** HIV **HRQOL ICF** 

**ICH IDMC** iDOR

IGF1R ILD

iORR iPFS **IRB IRC** 

IUD KD KL-6

v-Ki-ras2 Kirsten rat sarcoma viral oncogene homologue **KRAS** 

lactate dehydrogenase LDH

Medical Dictionary for Regulatory Activities MedDRA Ministry of Health, Labour and Welfare **MHLW** 

Medicines and Healthcare products Regulatory Agency **MHRA** 

MRI magnetic resonance imaging

NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events

NGS next-generation sequencing **NSCLC** non-small cell lung cancer objective response rate

overall survival progressive disease progression-free survival PK pharmacokinetic(s)

**PMDA** Pharmaceuticals and Medical Devices Agency of Japan

PP per-protocol PR partial response **PRO** patient-reported outcome

QD once daily

QLQ Quality of Life Questionnaire

QOL quality of life

QTc heart rate-corrected QT interval (calculated) QTcF corrected QT interval by the Fridericia formula RECIST Response Evaluation Criteria in Solid Tumors

ROS1 c-ros oncogene 1 SAE serious adverse event SAP statistical analysis plan

SD stable disease

sum of the longest diameters SLD

sum of the longest diameters
symptoms standardized Medical Dictionary for Regulatory Activities query **SMQ** 

SP-D surfactant protein-D

 $SpO_2$ percutaneous oxygen saturation **SRS** stereotactic radiosurgery

suspected unexpected serious adverse reaction **SUSAR** 

**TEAE** treatment-emergent adverse event

TKI tyrosine kinase inhibitor time of first occurrence of Cmax  $t_{\text{max}}$ upper limit of the normal range ULN

US **United States** 

Property of Fakeda. whole brain radiation therapy **WBRT** World Health Organization

### 4.0 OBJECTIVES

# 4.1 Primary Objectives

The primary objective is to evaluate efficacy of brigatinib in Japanese patients with ALK-positive advanced NSCLC.

- ORR will be evaluated in the refractory patients.
- PFS rate at 12 months in Kaplan-Meier plots (12 months PFS rate) will be evaluated in the TKI-naïve patients.

# 4.2 Secondary Objectives

The secondary objectives are:

- To confirm the clinical dose in Japanese patients.
- To characterize the efficacy of brigatinib as shown by following parameters
   For all enrolled patients (including TKI-naïve patients); DOR, PFS, disease control rate
   (DCR), time to response, and overall survival (OS).
   For the TKI-naïve patients: ORR
- To characterize the intracranial efficacy of brigatinib, as evidenced by iORR, duration of
  intracranial response (iDOR), and iPFS in patients with intracranial disease at baseline, from
  refractory and TKI-naïve cohorts.
- To assess patient-reported outcomes (PROs) of health-related quality of life (HRQOL) and symptoms of lung cancer with the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 (version 3.0), its lung cancer module QLQ-LC13, and the 5-level version of the EuroQol 5-dimensional questionnaire (EQ-5D-5L).
- To characterize the PK of brigatinib in Japanese patients.

# 4.3 Safety Objectives

The safety objective is to assess the safety and tolerability of brigatinib.

#### 4.4

# 4.5 Study Design

This is a nonrandomized, multicenter, phase 2, open-label study with a safety evaluation lead-in, to evaluate the efficacy and safety of brigatinib in Japanese patients with ALK-positive advanced NSCLC.

ns of Use The study consists of the safety evaluation lead-in part and the expansion part. The safety evaluation lead-in part allows patients with any line of prior ALK inhibitor which includes treatment-naïve patients; however, ALK inhibitor-naïve patients may be enrolled after the confirmation of first 3 DLT evaluable patients to have no more than 1 DLT during Cycle 1 by investigator's judgement. The expansion part consists of the TKI-naïve expansion cohort and the refractory expansion part, and the refractory expansion part includes the main cohort and & subcohort based on prior ALK inhibitor treatment. The TKI-naïve expansion cohort includes the patients who have not received any prior TKI including ALK inhibitor. In this cohort, the efficacy will be evaluated, and total of 32 patients will be enrolled. The main cohort of the refractory expansion part includes patients who had previously received alectinib (as their only ALK inhibitor) or both alectinib and crizotinib (regardless the sequence of those 2 ALK inhibitors). The main cohort of the refractory expansion part will be used for the primary analysis of efficacy, and a total of 47 patients will be enrolled in the main cohort of the refractory expansion part. Patients with all other sequences of up to 2 prior ALK inhibitor(s) may be included in the subcohort of the refractory expansion part. Such other ALK inhibitors include (1) crizotinib only, (2) ceritinib only, (3) lorlatinib only, (4) both crizotinib and ceritinib, (5) both alectinib and ceritinib, (6) both crizotinib and lorlatinib, (7) both alectinib and lorlatinib, and (8) both ceritinib and Iorlatinib. Up to 20 patients will be enrolled in the subcohort of the refractory expansion part.

In this study, brigatinib will be administered at 90 mg QD for the first 7 days and then 180 mg QD (90 mg QD  $\rightarrow$  180 mg QD). In the safety evaluation lead-in part, patients will be monitored for intensive PK, and the tolerability of 90 mg QD→180 mg QD dosing will be confirmed. If the 90 mg QD→180 mg QD dosing regimen is considered tolerable, additional patients enrolled in the expansion part will be treated with the same dosing schedule (90 mg OD→180 mg OD).

For the TKI-naïve expansion cohort, 32 patients will be enrolled and 12 month PFS rate will be evaluated as the primary endpoint. The primary analysis will be performed at around 10 months after the enrollment of the last subject in TKI-naïve expansion cohort. The sample size and evaluation timing may be adjusted based on results of second interim analysis of ALTA-1L study, and actual enrollment period of the TKI-naïve expansion cohort.

For the main cohort of the refractory expansion part, there are 2 stages: the first 29 patients in the main cohort are included in Stage 1, and further patients will be continuously enrolled into Stage 2. An interim analysis for futility and efficacy will be performed in the Stage 1 population when the first 29 post-alectinib patients have had the opportunity to complete at least 3 postbaseline scans (ie, after the Cycle 7 Day 1 disease assessment). Enrollment will not be suspended during evaluation of those 29 patients.

Following the screening period, eligible patients will be enrolled and treated with brigatinib. A patient is considered to be enrolled in the study when the first dose of brigatinib is administered.

Toxicity will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03, effective date 14 June 2010.

Response evaluation per RECIST version 1.1 will be done by both the investigator and an IRC. The primary analysis will performed on the results from the IRC.

Patients will be treated until they experience objective progressive disease (PD) per RECIST version 1.1, as assessed by the investigator, intolerable toxicity, withdrawal of consent, or discontinuation for any other reason. Treatment of patients with brigatinib may be continued at the tolerated dose level, despite investigator-assessed PD by RECIST version 1.1, if the patient otherwise has evidence of ongoing clinical benefit. In this case, discussions and agreements between the investigator and the sponsor's project clinician (or designee) are required.





# Safety Evaluation Lead-in Part

Nine DLT-evaluable patients will be enrolled in the safety evaluation lead-in part. The patients in the safety evaluation lead-in part will be hospitalized during Cycle 1 in general, and their condition will be closely monitored for safety and tolerability. Serial blood samples will be collected for the intensive PK profile. If a patient wishes to return home temporarily and the investigator confirms that the patient's symptoms are stable per the available data, then the patient may return home temporarily except on Days 1 through 10 and Days 22 and 23, provided this does not interfere with the study assessments. The investigator must document the confirmation record for stabilization of the patient's symptoms per the available data in an appropriate source record (eg, medical records) before the patient's temporary leave.

DLTs are defined in Section 8.2. Tolerability of the 90 mg QD—180 mg QD schedule will be determined on the basis of the DLTs observed in Cycle 1. If a DLT is observed in fewer than 3 of the 9 DLT-evaluable patients in the safety evaluation lead-in part the color QD regimen will be used for the patients enrolled.

# Expansion Part (Refractory Expansion Part and TKI-Naïve Expansion Cohort)

Patients in the refractory expansion part and the TKI-naïve expansion cohort may be managed on an outpatient basis, and the number of study sites will be increased up to approximately 40. Patients in the refractory expansion part and the TKI-naïve expansion cohort will undergo lessintensive PK blood sampling than patients in the safety evaluation lead-in part.

On an outpatient basis, patients will visit the hospital on Days 1, 8, and 15 of Cycle 1, and then on Day 1 of each cycle after Cycle 2. Tumor assessment will be performed every 2 cycles from Cycle 3 Day 1 through Cycle 15 Day 1, then every 3 cycles thereafter until the last dose of study drug. For patients who discontinue study treatment in the absence of PD, additional tumor assessment should continue at the same time points as the study treatment until PD or the start of another systemic anticancer therapy.

#### 5.0 **ANALYSIS ENDPOINTS**

#### 5.1 **Primary Endpoint**

The primary endpoints are:

- Confirmed ORR as assessed by an IRC, per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 in the main cohort of the refractory expansion part
- 12 months PFS rate as assessed by an IRC, per RECIST version 1.1 in the TKI-naïve expansion cohort

#### **Secondary Endpoints** 5.2

The secondary endpoints are:

- a) Efficacy endpoint in the TKI-naïve expansion cohort, the overall population of the refractory expansion part, and the safety evaluation lead-in part:
- Confirmed ORR, as assessed by an IRC, per RECIST version 1.1.
- b) Efficacy endpoints in the TKI-naïve expansion cohort, the main cohort of the refractory expansion part, the overall population of the refractory expansion part:
- DOR, as assessed by an IRC, per RECIST version 1.1.
- PFS, as assessed by an IRC, per RECIST version 1.1.

- DCR, as assessed by an IRC, per RECIST version 1.1.
- Time to response, as assessed by an IRC, per RECIST version 1.1.
- OS.
- CNS response, as assessed by IRC, per modified RECIST version 1.1 for assessment of
  intracranial efficacy (Appendix H) (iORR and iDOR in patients who had measurable
  CNS metastases, and iPFS in all patients).
- Time on treatment.
- c) Efficacy endpoints in the TKI-naïve expansion cohort, the main cohort of the refractory expansion part, and the safety evaluation lead-in part:
- Confirmed ORR, as assessed by the investigator, per RECIST version 1.1.
- PROs of HRQOL scores and symptoms of lung cancer, assessed with the EORTC QLQ-C30 (version 3.0), its lung cancer module QLQ-LC13, and the EQ-5D-5L (except for the safety evaluation lead-in part).
- d) PK endpoint in the safety evaluation lead-in part:
  - Brigatinib maximum observed plasma concentration (C<sub>max</sub>), time of first occurrence of C<sub>max</sub> (t<sub>max</sub>), and area under the plasma concentration-time curve (AUC) on Cycle 1 Days 1 and 22.

# 5.3 Safety Endpoints

The safety endpoints are:

- The number and percentage of patients with TEAEs in the overall population.
- The number and percentage of patients with Grade 3 or higher TEAEs in the overall population.
- The number and percentage of patients with serious TEAEs in the overall population.
- The number and percentage of patients discontinuing study drug because of TEAEs in the overall population.
- The number of patients with DLTs during Cycle 1 in the safety evaluation lead-in part.





# 6.0 DETERMINATION OF SAMPLE SIZE

The purpose of this phase 2 study is to determine efficacy of brigatinib in patients with ALK-positive NSCLC.

In the safety evaluation lead-in part, 9 DLT-evaluable patients will be enrolled for intensive safety and PK monitoring. This number of patients was derived from the following considerations: The meaningful intensive PK characterization needs to be conducted with more than 6 patients. It is assumed that 9 patients may be reasonable to secure the number of patients needed for intensive PK characterization, even with potential dropouts, and to evaluate the tolerability of the study drug. Also, 9 DLT-evaluable patients is enough to evaluate tolerability before expanding the dose cohort to a larger population using a conventional 3+3 design.

The sample size in the main cohort of the refractory expansion part was determined to allow confirmation that the true ORR (expected response rate) is greater than the threshold response rate of 15% for patients previously treated with alectinib alone and those treated with both alectinib and crizotinib. The rationale for the 15% response rate for the alectinib (with or without crizotinib) pretreated population is based on the consideration that compared with crizotinib, patients who have failed alectinib are less likely to respond to subsequent therapy because of alectinib's greater potency and better coverage of ALK mutations compared with crizotinib.

A sample size of 47 patients in the post-alectinib population of the refractory expansion part with the stopping rule mentioned in Section 13.2 will allow the study to have more than 90% power to rule out a threshold response rate when the true ORR is expected or higher than 35% with a 1-sided alpha of 0.025, according to the H1-minimax design in Englert [16].

The number of patients in the subcohort of the refractory expansion part (ie, patients previously treated with crizotinib only, ceritinib only, lorlatinib only, both crizotinib and ceritinib, both alectinib and ceritinib, both crizotinib and lorlatinib, or both ceritinib and lorlatinib) will be limited to 20. These patients will be included in evaluations of the overall population.

The sample size in the TKI-naïve expansion cohort was determined to allow confirmation that the true 12 months PFS rate (expected response rate) is greater than the threshold of 42.6% (estimated PFS rate at 12 months in Kaplan-Meier plots observed in ALTA-1L Crizotinib arm) for TKI-naïve patients.

A sample size of 32 patients in the TKI-naïve expansion cohort will allow the study to have approximately 80% power to rule out the threshold rate (42.6%) when the true 12 months PFS rate is expected or higher than 66.5% (estimated PFS rate at 12 months in Kaplan-Meier plots observed in ALTA-1L Brigatinib arm) with a 1-sided alpha of 0.05, considering 10% patients will discontinue the study follow-up before the 12 months milestone due to reasons other than disease progression assessed by IRC or death, and 8 months enrollment period. The primary

APPlicable Terms of Use analysis will be performed at around 10 months after the enrollment of the last subject in the TKI-naïve expansion cohort. The sample size and evaluation timing may be adjusted based on results of second interim analysis of ALTA-1L study, and actual enrollment period of the TKInaïve expansion cohort.

Overall, the total number of patients will be approximately 110 patients.

#### 7.0 METHODS OF ANALYSIS AND PRESENTATION

#### 7.1 **General Principles**

All statistical analyses will be conducted using SAS® Version 9.4, or higher.

A statistical test for the primary endpoint will be reported as 1-sided and will be assessed at  $\alpha$ =0.025 significance level and all confidence intervals will be reported as 2-sided unless otherwise stated. P-values will be rounded to 4 decimal places prior to assessment of statistical significance.

Means and medians will be presented to 1 more decimal place than the recorded data. The standard deviations (SDs) will be presented to 2 more decimal places than the recorded data. Confidence intervals about a parameter estimate will be presented using the same number of decimal places as the parameter estimate.

Where appropriate, variables will be summarized descriptively by study visit. For the categorical variables, the count and proportions of each possible value will be tabulated. The denominator for the proportion will be based on the number of subjects who provided non-missing responses to the categorical variable. For continuous variables, the number of subjects with non-missing values, mean, median, SD, minimum, and maximum values will be tabulated.

#### **Study Definitions** 7.1.1

How to convert a time-to-event endpoint unit from day to month:

value (Month)= value (Day)/30.4375

Dose intensity:

Total amount of doses taken/(Last non-zero dose date – First dose date +1)

Relative Dose Intensity:

(Total amount of dose taken /Total amount of dose planned per initial dose)\*100

Objective Response Rate(ORR):

The proportion of patients who are confirmed to have achieved CR or PR

Confirmed responses

Responses that persist on repeat imaging 4 weeks (allowing a minus 3-day time window) or more after initial response, which will be confirmed by the investigator or IRC.

# Duration of Response(DOR):

The time between the first documentation of objective tumor response (CR or PR) and the first subsequent documentation of objective PD or death due to any cause, whichever occurs first

# Progression-Free Survival (PFS):

The time from the start of study treatment to the first documentation of objective PD or to death due to any cause, whichever occurs first.

- Based only on radiological assessments verified by an IRC. Clinical progression is not considered a progression endpoint.
- The date of death when the patient is closely followed. However, deaths occurring after two or more missed visits are censored at the last visit
- The detailed scheme of progression and censoring for the primary analysis of PFS is specified in Table 7.a.

Table 7.a The Scheme of Progression and Censoring for PFS

| Situation | Date of progression or censoring | Outcome |
|---|---|---|
| Documented disease progression or | Earliest of the following: | Progressed |
| death with no baseline disease assessment | Date of death | |
| assessment | Date of progression | |
| New anticancer treatment (including palliative radiotherapy and cancer- | Date of last adequate radiological assessment prior to initiation of new anticancer treatment | Censored |
| related surgery) started prior to | (including palliative radiotherapy and cancer- | |
| documented disease progression or | related surgery) | |
| death | (O' | |
| Death or PD without more than 1 | Date of death or first PD whichever occurred | Progressed |
| missing radiographic assessment | first | |
| Death or PD after two or more missing | Date of last adequate radiological assessment | Censored |
| radiographic assessments | | |
| No progression or death | Date of last adequate radiological assessment | Censored |

# Disease Control Rate (DCR):

The proportion of patients who are confirmed to have achieved CR or PR or have a best overall response of stable disease (SD) for 6 weeks or more after initiation of study drug.

# Time to response:

The time interval from the date of the first dose of study treatment until the initial observation of CR or PR for patients with confirmed CR/PR.

# Overall Survival (OS):

The time from the start of study treatment to the date of death.

Best response in target lesions:

The maximum unsigned decrease (or the minimum increase if no decrease) in percentage in the sum of the longest dimensions of the target lesions at a single assessment as compared with baseline.

Time on treatment

Time on treatment is defined as the time interval from the first dose to the last dose of assigned study treatment.

ILD/Pneumonitis Events:

The search strategy included manual selection of PTs of Interstitial lung disease and Pneumonitis.

Bradycardia Events:

The search strategy included manual selection of PTs of Ibradycardia, Central bradycardia, Heart rate decreased, Sinus bradycardia, Bradyarrhythmia, Atrioventricular block, Atrioventricular block complete, Atrioventricular block first degree and Atrioventricular block second degree.

Hypertension Events:

The search strategy included manual selection of PTs of Accelerated hypertension, Blood pressure diastolic increased, Blood pressure increased, Blood pressure systolic increased, Diastolic hypertension, Hypertension and Systolic hypertension.

GI Events:

Some PTs were retrieved manualy from SMQ; Gastrointestinal nonspecific symptoms and therapeutic procedures. For other GI events, the search strategy included manual selection of PTs of Dysphagia, Gastrointestinal tract irritation, Regurgitation, Retching and Vomiting projectile. Further details are given in Appendix 2.

Increased Insulin/ Hyperglycemia Events:

Hyperglycemia Events. The search strategy included manual selection of PTs of Blood glucose increased, Diabetes mellitus, Glycosylated haemoglobin increased, Hyperglycaemia, Insulin resistant diabetes, Insulin-requiring type 2 diabetes mellitus, Type 1 diabetes mellitus, Type 2 diabetes mellitus and Type 3 diabetes mellitus.

Increased Insulin Events: The search strategy included manual selection of PTs of Blood Insulin increased and Hyperinsulinaemia.

Hyperglycemia Events and Increased Insulin Events were analyzed and tabulated together.

Hepatic Events

Some PTs were retrieved manualy from SMQ; Liver related investigations, signs and symptoms, Cholestasis and jaundice of hepatic origin, Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions and Hepatitis, non-infectious. Further details are given in Appendix 2.

## **Elevated CPK**

The search strategy included manual selection of PTs of Blood creatine increased, Blood creatine phosphokinase increased, Hypercreatinaemia, Blood creatine phosphokinase MB increased, Blood creatine phosphokinase BB increased,

# Muscle Toxicity

The search strategy included manual selection of PTs of Muscle necrosis, Myoglobin blood increased, Myoglobin blood present, Myoglobin urine present, Myoglobinaemia, Myoglobinuria, Myopathy, Myopathy toxic, Necrotising myositis, Rhabdomyolysis, Biopsy muscle abnormal, Muscle discomfort, Muscle disorder, Muscle fatigue, Muscular weakness, Musculoskeletal discomfort, Musculoskeletal disorder, Musculoskeletal pain, Myalgia, Myositis and Musculoskeletal chest pain.

#### **Pancreatic Events**

Chemical Pancreatitis: The search strategy included manual selection of PTs of Amylase abnormal, Amylase increased, Hyperamylasaemia, Hyperlipasaemia, Lipase abnormal, Lipase increased, Pancreatic enzyme abnormality, Pancreatic enzymes abnormal, Pancreatic enzymes increased and Ultrasound pancreas abnormal.

Clinical Pancreatitis: The search strategy included manual selection of PTs of Haemorrhagic necrotic pancreatitis, Ischaemic pancreatitis, Oedematous pancreatitis, Pancreatic abscess, Pancreatic haemorrhage, Pancreatic necrosis, Pancreatitis, Pancreatitis acute, Pancreatitis haemorrhagic, Pancreatitis necrotising and Pancreatitis relapsing.

Chemical and clinical pancreatic events were analyzed and tabulated together.

# Peripheral Neuropathy Events

A broad search strategy was used for the retrieval of all active PTs from the SMQ: Peripheral neuropathy.

# Skin and Subcutaneous Events

The search strategy was used for the retrieval of all active PTs from the SOC; Skin and Subcutaneous Events.

# Visual Impairment Events

The search strategy was used for the retrieval of all active PTs from the HLGT; vision disorder, some PTs were retrieved from SMQs; retinal disorder, glaucoma, lens disorder. For other Visual Impairment events, the search strategy included manual selection of PTs. Further details are given in Appendix 2.

# Photosensitivity

The search strategy was used for the retrieval of all active PTs from the HLT; photosensitivity and photodermatosis conditions. Further details are given in Appendix 2.

CNS involvement at Screening:

The subjects with Brain and Leptomeningeal Involvement at Screening

Treatment-Emergent Adverse Events leading to study drug dose modification:

TEAE leading to dose discontinuation, dose interruption, or dose reduction

The subject who administrated any Chemo therapy:

and subject to the app The subjects who administrated the medication whose code are matched in the following table as prior anticancer therapy

| 1 5 |
|--------------------------------------|
| Bevacizumab |
| Carboplatin |
| Chemotherapeutics |
| Cisplatin |
| Docetaxel |
| Gimeracil;Oteracil potassium;Tegafur |
| Gimeracil;Oteracil;Tegafur |
| Motesanib |
| Nivolumab |
| Paclitaxel |
| Pembrolizumab |
| Pemetrexed disodium |
| Tegafur;Uracil |
| Vinorelbine tartrate |

#### **Definition of Study Days** 7.1.2

Study Day 1 is defined as the date on which a subject is administered their first dose of the medication. Other study days are defined relative to the Study Day 1 with Day 1 being Study Day 1 and Day -1 being the day prior to Study Day 1.

#### **Definition of Study Visit Windows** 7.1.3

For each visit, observation obtained in the corresponding time interval will be used. If more than one observation lies within the same visit window, the observation with the closest Day to the scheduled Day will be used. If there are two observations equidistant to the scheduled Day, the later observation will be used.

# HRQOL scores(EORTC QLQ-C30, QLQ-LC13, and EQ-5D-5L), 12-lead ECG, ECOG performance status, and Testosterone

| | Scheduled Day<br>(days) | Time Interval (days) | |
|---|---|---|---|
| Visit | | Day* | Follow-up Day |
| Baseline | Day from first visit in cycle1: | 1 | -14 - 1 |
| Cycle 2 | Day from first visit in cycle2: | 1 | -3 - 29 |
| Cycle 3 | Day from first visit in cycle3: | 1 | -3 - 29 |
| Cycle 4 | Day from first visit in cycle4: | 1 | -3 - 29 |
| Cycle 5 | Day from first visit in cycle5: | 1 0 | -3 - 29 |
| Cycle 6 and beyond | Day from first visit in each cycle: | 1 (2) | -3 - 29 |

<sup>\* &</sup>quot;Day" indicates day after first visit in cycle which is mentioned in "Scheduled Study Day".

If the data is in the scope of several visits, the data will be regarded as the candidate data of the latest visit.

# <u>Laboratory Assessments except HbA1c and Testosterone</u>

| | Scheduled Day | Time | Time Interval (days) |
|---|---|---|---|
| Visit | (days) | Day* | Follow-up Day |
| Baseline | Day from first visit in cycle1: | 1 | -14 - 1 |
| Cycle 1 Day15 | Day from first visit in cycle1: | 15 | 2 - 29 |
| Cycle 2 | Day from first visit in cycle2: | 1 | -3 - 29 |
| Cycle 3 | Day from first visit in cycle3: | 1 | -3 - 29 |
| Cycle 4 | Day from first visit in cycle4: | 1 | -3 - 29 |
| Cycle 5 | Day from first visit in cycle5: | 1 | -3 - 29 |
| Cycle 6 and beyond | Day from first visit in each cycle: | 1 | -3 - 29 |

<sup>\* &</sup>quot;Day" indicates day after first visit in cycle which is mentioned in "Scheduled Study Day".

If the data is in the scope of several visits, the data will be regarded as the candidate data of the latest visit.

# Vital signs

| | Scheduled Day | Time Interval (days) | |
|---|---|---|---|
| Visit | (days) | Day* | Follow-up Day |
| Basetine | Day from first visit in cycle1: | 1 | -14 - 1 |
| Cycle I Day8 | Day from first visit in cycle1: | 8 | 2 - 11 |
| Cycle 1 Day15 | Day from first visit in cycle1: | 15 | 12 - 29 |
| Cycle 2 | Day from first visit in cycle2: | 1 | -3 - 29 |
| Cycle 3 | Day from first visit in cycle3: | 1 | -3 - 29 |
| Cycle 4 | Day from first visit in cycle4: | 1 | -3 - 29 |
| Cycle 5 | Day from first visit in cycle5: | 1 | -3 - 29 |
| Cycle 6 and beyond | Day from first visit in each cycle: | 1 | -3 - 29 |

<sup>\* &</sup>quot;Day" indicates day after first visit in cycle which is mentioned in "Scheduled Study Day".

If the data is in the scope of several visits, the data will be regarded as the candidate data of the latest visit.

# HbA1c

| | Scheduled Day | Time | Interval (days) |
|---|---|---|---|
| Visit | (days) | Day* | Follow-up Day |
| Baseline | Day from first visit in cycle1: | 1 | -14 - 1 |
| Cycle 4 and beyond | Day from first visit in each cycle: | 1 | -3 - 29 |

<sup>\* &</sup>quot;Day" indicates day after first visit in cycle which is mentioned in "Scheduled Study Day".

If the data is in the scope of several visits, the data will be regarded as the candidate data of the latest visit.

# 7.1.4 Methods for Handling Missing Data and Specific Data

All available efficacy and safety data will be included in data listing and tabulations. No imputation of values for missing data will be performed unless otherwise specified.

- For ORR as assessed by an IRC, if any tumor response of post baseline is not assessed or any tumor response of baseline is not confirmed as measurable disease per the IRC, the patients will be treated as the one who are <u>not</u> confirmed to have achieved CR or PR
- For ORR as assessed by an investigator, if any tumor response of post baseline is not assessed or any tumor response of baseline is not confirmed as measurable disease per the investigator, the patients will be treated as the one who are <u>not</u> confirmed to have achieved CR or PR
- For DCR, patients with only non-measurable disease who had a CR or non-CR/non-PD will be considered as having achieved DCR.
- For DOR, if tumor response cannot be confirmed, the patient will not be analyzed.
- For EORTC QLQ-C30, QLQ-LC13, published scoring manuals and guidelines will be used to calculate scores and handle missing data.
- For stage at Screening, if no data has been input in CRF, the stage at initial diagnosis will be used as the stage at screening,
- For clinical laboratory tests, values less than the lower limit of quantification will be treated as value of lower limit when calculating the descriptive statistics.
- Disease duration with first diagnosis date of ALK + non small cell lung cancer that are completely or partially missing will be derived as follows:
  - If the year is missing, then the disease duration will be treated as missing.
  - If the year is present but the month is missing, then the month will be treated as January for the calculation.

# 7.2 Analysis Sets

The refractory expansion part and safety evaluation lead-in part:

Safety population will be defined as patients who receive at least 1 dose of study drug will be used for all safety analyses.

Full analysis set (FAS) population will be defined as all patients who receive at least 1 dose of study drug.

FAS-P population, the main analysis set used for primary efficacy analysis, will be defined a subset of the FAS population consisting of first 47 patients in the main cohort of the expansion part.

Per-protocol (PP) population will be defined as a subset of the FAS-P population including patients who do not have a major protocol violation listed below:

- Subjects who did not meet inclusion criteria #3, #4, #6 or, #10.
- Subjects who met exclusion criteria #9, #10, #11, #13 or, #14.
- Subjects who have violated the following rules specified in section 8.5.
  - Any other systemic anticancer therapy including, but not limited to, chemotherapeutic
    agents, immunotherapy, biological response modifiers (excluding growth factors),
    radiotherapy, and/or systemic hormonal therapy (with the exception of local therapies,
    such as SRS and WBRT, used for palliative or symptomatic control of existing lesions,
    with appropriate treatment interruption at the discretion of the investigator). Hormonal
    contraception is allowed.
  - Use of any other investigational drug or device.
  - Extensive surgery requiring in-patient care (patients may have an interruption in therapy for 14 days should emergency surgery be required).

PK population will be defined as patients with sufficient dosing and PK data to reliably estimate PK parameters as determined by the clinical pharmacologist

DLT population will be a subset of the DLT evaluable subject who completes at least 75% of planned cumulative doses in safety evaluation lead-in part.

The TKI-naïve expansion cohort:

Safety population will be defined as patients who receive at least 1 dose of study drug will be used for all safety analyses.

Full analysis set (FAS) population will be defined as all patients who receive at least 1 dose of study drug.

PK population will be defined as patients with sufficient dosing and PK data to reliably estimate PK parameters as determined by the clinical pharmacologist

Per-protocol (PP) population will be defined as a subset of the FAS population including patients who do not have a major protocol violation listed below:

• Subjects who did not meet inclusion criteria #3, #4, #6 or, #10.

- Subjects who met exclusion criteria #1, #9, #10, #11, #13 or, #14.
- Subjects who have violated the following rules specified in section 8.5.
  - Any other systemic anticancer therapy including, but not limited to, chemotherapeutic
    agents, immunotherapy, biological response modifiers (excluding growth factors),
    radiotherapy, and/or systemic hormonal therapy (with the exception of local therapies,
    such as SRS and WBRT, used for palliative or symptomatic control of existing lesions,
    with appropriate treatment interruption at the discretion of the investigator). Hormonal
    contraception is allowed.
  - Use of any other investigational drug or device.
  - Extensive surgery requiring in-patient care (patients may have an interruption in therapy for 14 days should emergency surgery be required).

# 7.3 Disposition of Subjects

# 7.3.1 Study Information

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis

Variable(s): Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit

MedDRA Version

WHO Drug Version

SAS Version Used for Creating the Datasets

Analytical

Method(s):

(1) Study Information

Study information shown in the analysis variables section will be provided.

# 7.3.2 Screen Failures

Analysis Set: All Subjects Who Did Not Enter the Treatment Period

Analysis

Variable(s): Age (years) [20<= - <65, 65<= - <=Max]

[20<= - <50, 50<= - <65, 65<= -

<75,75<=-<=Max]

Gender [Male, Female]

Analytical Method(s):

(1) Screen Failures

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

# 7.3.3 Subject Eligibility

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis

Variable(s): Eligibility Status [Eligible for Entrance into the

Treatment Period, Not Eligible for

Entrance into the Treatment

Period]

Primary Reason for Subject Not

Being Eligible

[Adverse Event, Death, Lost to Follow-up, Protocol Deviation, Screen Failure, Study Terminated

by Sponsor, Withdrawal by

Subject, Other]

Analytical

Method(s):

(1) Eligibility for Entrance into the Treatment Period

Frequency distributions will be provided. When calculating percentages for the primary reasons for subject not being eligible, the total number of

ineligible subjects will be used as the denominator.

# 7.3.4 Number of Subjects Who Entered the Treatment Period by Site

Analysis Set: All Subjects Who Entered the Treatment Period

**Analysis** 

Variable(s): Status of Entrance into the

[Entered]

**Treatment Period** 

Stratum: Site

[Site name and number will be used

as categories]

Analytical Method(s):

(1) Number of Subjects Who Entered the Treatment Period by Site

Frequency distribution will be provided for each stratum.

# 7.3.5 Disposition of Subjects

Analysis Set: All Subjects Who Entered the Treatment Period

All Subjects Who Entered the Treatment Period in the main cohort

Analysis

Variable(s): Subject Status(End of Treatment) [Completed, Adverse Event, Death,

Lost to Follow-up, Progressive Disease, Protocol Deviation, Study Terminated by Sponsor,

Symptomatic Deterioration, Withdrawal by Subject, Other,

Ongoing]

Subject Status(Follow-up) [Death, Lost to Follow-up, Study

Terminated by Sponsor, Withdrawal by Subject, Other,

Ongoing]

Analytical Method(s):

(1) Disposition of Subjects

Frequency distributions will be provided. When calculating percentages for the reasons for not being treated, the total number of subjects not treated by the study drug will be used as the denominator. When calculating percentages for the reasons for discontinuation, the total number of subjects who prematurely discontinued will be used as the denominator.

Protocol Deviations

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis

7.3.6

Variable(s): Protocol Deviation [Entry Criteria, Concomitant Medication,

Procedure Not Performed Per Protocol(Primary Endpoint or Safety Related), Study Medication, Withdrawal Criteria, Major GCP Violations]

Analytical Method(s):

(1) Protocol Deviations

Frequency distribution will be provided for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the same category will be counted only once.

#### 7.3.7 **Analysis Sets**

Analysis Set: All Subjects Who Entered the Treatment Period

All Subjects Who Entered the Treatment Period in the main cohort

(For the refractory patients)

All Subjects Who Entered the Treatment Period in the safety evaluation

lead-in part. (For the refractory patients)

**Analysis** 

Variable(s): [Categories are based on Subject Handling of Subjects

Evaluability List]

**Analysis Sets** 

Full Analysis Set [Included]

Full Analysis Set P [Included]

(For the refractory patients)

Per Protocol Set [Included]

Safety Analysis Set [Included]

PK population [Included]

DLT population [Included]

(For the refractory patients

Analytical Method(s):

(1) Subjects Excluded from Analysis Sets

(2) Analysis Sets

For DLT population, frequency distributions will be provided for the subjects in the safety evaluation lead-in part. For other populations, it will be done in overall population and main cohort. For (1), a subject who has several reasons for exclusion will be counted once in each appropriate category for each analysis set. A subject who has several reasons for exclusion that can be classified into the same category will be counted only once.

For analysis on Full Analysis Set P, all subjects who entered the treatment period in the main cohort will be used as analysis set.

# **Demographic and Other Baseline Characteristics**

Analysis Set: Safety analysis set

Full Analysis Set

# Full Analysis Set P(For the refractory patients)

| . 1 | |
|----------|-----------------------------------------|
| Ana | VS1S |
| 1 111111 | , ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, |

Variable(s):

 $[20 \le - <65, 65 \le - <= Max]$ Age (years)

[20<= - <50, 50<= - <65, 65<= -

<75,75<=-<=Max

Gender [Male, Female]

[Min<= - <150, 150<= - <160, 160<= - <170, 170<= - <= Max] Height (cm)

[Min<= - <50, 50<= <60, Weight (kg) at Baseline

60<= - <70, 70<=

**Smoking Classification** The subject has never smoked,

> The subject is a current smoker, The subject is an ex-smoker]

[IA, IB, IIA, IIB, IIIA, IIIB, IIIC, Stage at Initial Diagnosis

JV, Unknown or not staged]

[IA, IB, IIA, IIB, IIIA, IIIB, IIIC, Stage at Screening

IV, Unknown or not staged,

Refractory, Other]

Histopathological Classification of

**NSCLC** 

[Adenocarcinoma, Adenosquamous

carcinoma, Large cell, Squamous,

Unknown, Other]

Lung involvement at Screening [Left Lung, Right Lung, Both

Lungs, Lungs not involved]

CNS involvement at Screening [Yes, No]

Property of Takedai Time from Initial Diagnosis to study treatment (months)

**ECOG Performance Status** [0, 1, 2, 3, 4]

Was the genetic status of ALK in

tumor tissue assessed? [Yes, No]

ALK mutation method of

assessment

FISH-Vysis

[Yes] FISH-non Vysis [Yes]

| Brigatinib-2001<br>Statistical Analysis Plan Amendment 6 | Page 28 of 83<br>13 Jul 2021 |
|---|---|
| Vysis ALK Break Apart FISH<br>Probe Kit | [Yes] |
| Nichirei Histofine RALK iAEP<br>Kit | TY 1 |
| Ventana ALK (D5F3) CDx<br>Assay | [Yes] |
| RT-PCR | [Yes] |
| Sequencing | [Yes] |
| Unknown | [Yes] |
| Other | [Yes] |
| | [Yes] |
| Was an abnormality detected? | [Yes, No, Unknown] |
| fusion partner | [EML4, TFG, KIF5B, NPM,<br>Fusion partner unknown, Other<br>fusion partner] |
| ALK secondary mutation | H |
| T1151Tins L1152R C1156Y I1171T I1171N | [Yes] |
| L1152R | [Yes] |
| C1156Y | [Yes] |
| I1171T | [Yes] |
| I1171N (11) | [Yes] |
| I1171S | [Yes] |
| F1174C | [Yes] |
| F1174L | [Yes] |
| V1180L | [Yes] |
| L1196M | [Yes] |
| L1198F | [Yes] |
| G1202R | [Yes] |
| G1202del | [Yes] |
| I11718<br>F1174C<br>F1174L<br>V1180L<br>L1196M<br>L1198F<br>G1202R<br>G1202del<br>D1203N<br>S1206Y | [Yes] |
| S1206Y | [Yes] |

E1210K [Yes] G1269A [Yes] Unknown [Yes] Other [Yes]

Any Anticancer Therapies [Yes, No]

[Alectinib only, Crizotinib and C Regimen

> Alectinib, Crizotinib only, Ceritinib only, Lorlatinib only, Crizotinib and Ceritinib. Alectinib and Ceritinib, Crizotinib and Lorlatinib, Alectinib and

Lorlatinib, Ceritinib and Lorlatinib,

Other]

Any Prior Chemo therapy Any Prior Radiotherapy

**Anatomic Site** 

Lung [Yes] Mediastinal Lymph Nodes [Yes] Bone [Yes] Brain [Yes] Other [Yes]

Analytical Method(s):

(1) Summary of Demographics and Baseline Characteristics Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

#### 7.5 **Medical History and Concurrent Medical Conditions**

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Medical History

**Concurrent Medical Conditions** 

Analytical

Method(s):

(1) Medical History by System Organ Class and Preferred Term

# (2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided. MedDRA dictionary will be used for coding. Summaries will be provided using SOC and PT, where SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

A subject with multiple occurrences of medical history or concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of medical history or concurrent medical condition within a PT will be counted only once in that PT.

# 37114 and subject to 7.6 **Medication History and Concomitant Medications**

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Medication History

Concomitant Medications

Analytical

Method(s):

- (1) Medication History by Preferred Medication Name
- (2) Concomitant Medications That Started Prior to and Were Ongoing at Baseline as well as Those That Started After Baseline by Preferred Medication Name

Frequency distributions will be provided. WHO Drug dictionary will be used for coding Summaries will be provided using preferred medication names and sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same preferred medication name will be counted only once for that preferred medication name.

#### 7.7 Study Drug Exposure and Compliance

Analysis Set: Safety Analysis Set

Safety Analysis Set in the main cohort

Analysis Variable(s):  $[0, 1, 2, 3, 4, 5, 6 \le - \le Max]$ Number of treated cycle

Total amount of doses taken (mg)

Dose intensity (mg/day)

Relative dose intensity (%)

Duration of treatment (month)

Duration of follow-up (month)

Analytical Method(s):

(1) Study Drug Exposure and Compliance

ave applicable terms of Use while the applicable terms of Use Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

#### 7.8 **Efficacy Analysis**

#### 7.8.1 **Primary Efficacy Endpoint(s)**

#### 7.8.1.1 Primary Analysis

Analysis Set: Full Analysis Set P(For the refractory patients)

Full Analysis Set (For TKI-naïve Patients)

**Analysis** 

Variable(s):

Confirmed ORR as assessed by an IRC(For the refractory patients)

PFS as assessed by an IRC (For TKI-naïve Patients)

Analytical

Method(s):

The point estimate and its 2-sided 95% confidence interval will be summarized. The point estimate will be calculated by the method suggested by Kunzmann(2017) with weight function of uniform distribution of [0,1], which means that the point estimate will  $((x_1+x_2+1)/49)x_100$ . X1 and x2 represents the number of events at IA for the first 29 patients in the main cohort and the number of events at PA for the last 18 patients in the main cohort, respectively.

The confidence interval will be done based on the Clopper-Pearson type.

For PFS, the rate at 12 and, 24 months and the associated two-sided 90% confidence intervals with complementary log-log link will also be provided using the Kaplan-Meier method.

7.8.1.2 Secondary Analysis

Analysis Set: Per Protocol Set(For the refractory patients)

Analysis

Variable(s): Confirmed ORR as assessed by an IRC

PFS as assessed by an IRC (For TKI-naïve Patients)

Analytical

Method(s): The point estimate and its 2-sided 95% confidence interval will be

summarized. The point estimate will be calculated based on maximum likelihood estimation. The confidence interval will be done based on the

Clopper-Pearson type.

For PFS, the rate at 12 and, 24 months and the associated two-sided 90%

confidence intervals with complementary log-log link will also be

provided using the Kaplan-Meier method.

# 7.8.2 Secondary Efficacy Endpoint(s)

7.8.2.1 Confirmed ORR by the investigator

Analysis Set: Full Analysis Set P(For the refractory patients)

**Analysis** 

Variable(s): Confirmed ORR as assessed by the investigator

Analytical

Method(s): The point estimate and its 2-sided 95% confidence interval will be

summarized. The point estimate will be calculated based on maximum likelihood estimation. The confidence interval will be done based on the

Clopper-Pearson type.

7.8.2.2 Confirmed ORR by an IRC

Analysis Set: Full Analysis Set

Full Analysis Set P(For the refractory patients)

**Analysis** 

Variable(s): Confirmed ORR as assessed by an IRC

Analytical Method(s):

The point estimate and its 2-sided 95% confidence interval will be summarized. The point estimate will be calculated based on maximum likelihood estimation. The confidence interval will be done based on the Clopper-Pearson type.

# 7.8.2.3 Other assessment by an IRC

Analysis Set: Full Analysis Set

Full Analysis Set P(For the refractory patients)

Patients who had measurable CNS metastases in Full Analysis Set

Patients who had measurable CNS metastases in Full Analysis Set P

(For the refractory patients)

Analysis Variable(s):

DOR as assessed by an IRC

PFS as assessed by an IRC(For the refractory patients)

DCR as assessed by an IRC

Time to response as assessed by an IRC

OS

CNS response

iORR by an IRC

iDOR by an IRC

iPFS by an IRC

Time to intracranial response as assessed by an IRC

Time on treatment

Best response in target lesions

Analytical Method(s):

For iDOR and DOR, the cumulative incidences and the two-sided 95% confidence intervals will be provided using the Kaplan-Meier method. For DOR, Time to response, and Time to intracranial response as assessed by an IRC, summary of descriptive analysis will be provided for subjects with confirmed CR or PR.

For Time on treatment, the summary of descriptive analysis will be provided and swimmer's plot will be presented.

For iPFS, PFS, and OS, the rate at 12 and, 24 months and the associated two-sided 95% confidence intervals with complementary log-log link will also be provided using the Kaplan-Meier method.

Especially, for iPFS, considering the progression by investigator assessment as competing risk and only intracranial progression by IRC as event, the cumulative incidence function for event will be provided.

Additionally, for the analysis for TKI-naïve patients, the same analysis mentioned above will be performed in Per Protocol Set.

For iORR, DCR, CNS response, the point estimate and its 2-sided 95% confidence interval will be summarized. The point estimate will be calculated based on maximum likelihood estimation. The confidence interval will be done based on the Clopper-Pearson type.

For iDOR and iORR, patients who had measurable CNS metastases in Full Analysis Set or in Full Analysis Set P will be used as analysis set.

For best response in target lesions, summary of descriptive analysis will be provided with a waterfall plot.

# 7.8.2.4 EORTC QLQ-C30

Analysis Set: Full Analysis Set in expansion part

Full Analysis Set P (For the refractory patients)

Analysis

Global health status

Variable(s):

Global health status

Functional scales

Physical functioning

Role functioning

Emotional functioning

Cognitive functioning

Social functioning

Symptom scales

Fatigue

Nausea and vomiting

Pain

Dyspnoea

Insomnia

Appetite loss Constipation Diarrhoea

Financial difficulties

Baseline, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6, Cycle 7, Cycle 8, Visit:

Cycle 9, Cycle 10, Cycle 11, Cycle 12, Cycle 13, Cycle 14, Cycle 15.

Cycle 16, Cycle 17, Cycle 18

Analytical

Method(s): Descriptive statistics for observed values for each visit and changes from ind subject

baseline will be provided.

7.8.2.5 EORTC QLQ-LC13

Analysis Set: Full Analysis Set in expansion part

Full Analysis Set P(For the refractory patients)

**Analysis** 

Variable(s):

Dyspnoea

Coughing

Haemoptysis

Sore mouth

Dysphagia (

Peripheral neuropathy

Alopecia

Pain in chest

Pain in arm or shoulder

Pain in other parts

Baseline, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6, Cycle 7, Cycle 8,

Cycle 9, Cycle 10, Cycle 11, Cycle 12, Cycle 13, Cycle 14, Cycle 15,

Cycle 16, Cycle 17, Cycle 18
Analytical

Method(s):

Only and subject to the applicable Terms of Use only and subject to the applicable Terms of Use Descriptive statistics for observed values for each visit and changes from

baseline will be provided.

7.8.2.6 *EQ-5D-5L* 

Analysis Set: Full Analysis Set in expansion part

Full Analysis Set P(For the refractory patients)

**Analysis** 

Variable(s): **Mobility** 

Selfcare

Activity

Pain

Anxiety

EQ VAS

Index Value

Baseline, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6, Cycle 7, Cycle 8, Visit:

Cycle 9, Cycle 10, Cycle 11, Cycle 12, Cycle 13, Cycle 14, Cycle 15,

Cycle 16, Cycle 17, Cycle 18

Analytical

Method(s): For categorical variables, frequency distributions for each visit will be

> provided. And for continuous variables, descriptive statistics for observed values for each visit and changes from baseline will be

provided.

7.8.3 Additional Efficacy Endpoint(s)

Confirmed ORR by an IRC by the previous ALK inhibitor regimen 7.8.3.1

Analysis Set: Full Analysis Set

Full Analysis Set-P(For the refractory patients)

Analysis

Variable(s): Confirmed ORR as assessed by an IRC (For the refractory patients)

PFS as assessed by an IRC (For TKI-naïve Patients)

Stratified

Variable(s): Age (years)  $[20 \le -.. \le 65, 65 \le -.. \le Max]$ 

Gender [Male, Female]

CNS involvement at Screening [Yes, No]

Previous ALK Inhibitor Regimen
(For the refractory patients)

[Alectinib only, Crizotinib and Alectinib, Crizotinib only, Ceritinib only, Lorlatinib only,

Crizotinib and Ceritinib, Alectinib

and Ceritinib, Other]

[Containing G1202R, Not

containing G1202R but containing

other, No or unknown somatic

mutation]

[Yes, No]

Any Prior Chemo Therapy

ALK secondary mutation

Analytical Method(s):

The point estimate and its 2-sided 95% confidence interval will be summarized by stratified variable. The point estimate will be calculated based on maximum likelihood estimation. The confidence interval will be done based on the Clopper-Pearson type.

For PFS, the rate at 12 and, 24 months and the associated two-sided 90% confidence intervals with complementary log-log link will also be provided using the Kaplan-Meier method by stratified variable.

## 7.8.3.2 Proportion of patients with event

Analysis Set: Full Analysis Set P (For the refractory patients)

Full Analysis Set

Analysis

Variable(s) Proportion of patients with PFS event

Proportion of patients with iPFS event (For the naive patients)

Proportion of patients with OS event Proportion of patients with DOR event Analytical Method(s): Lations of brigatinib and AP26123

A population

Plasma concentrations of brigatinib and AP26123

(Safety Evaluation Lead-in Part)

//isit: Cycle 1 Day 1 and Cycle 1 Day 22

redose and 0.5, 1, 2, 4, 6, 8, 12, 2"

te of morning dose at Day

it: Cycle 1 Day

le 4 Day

1

#### 7.9 Pharmacokinetic/Pharmacodynamic Analysis

#### 7.9.1 Pharmacokinetic Analysis

#### 7.9.1.1 Plasma concentrations of brigatinib and AP26123

Analysis Set: PK population

**Analysis** 

Variable(s):

Time Point:

Cycle 4 Day 1, Cycle 5 Day D

Predose

(Expansion Part)

Visit: Cycle 1 Day 1, Cycle 1 Day 8, and Cycle 1 Day 15

Predose and P-4 hours postdose (relative to start time of morning dose at

Day 1, 8, or 15)

Predose Predose Visit: Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1

## Analytical Method(s):

The following summaries will be provided for each analyte by analysis set.

- (1) Descriptive statistics (mean, standard deviation, minimum, median and maximum) for observed values will be provided for each time point by dose. In addition, %CV, geometric mean, and geometric %CV will be provided
- (2) Observed values will be plotted using individual case plot
- (3) Mean of plasma concentrations will be plotted by time point using linear scale.
- (4) Mean of plasma concentrations will be plotted by time point using common log scale.

## 7.9.1.2 Plasma PK parameters of brigatinib and AP26123

Analysis Set: PK population

Analysis

Variable(s):

Plasma Concentrations of brigatinib and AP26123

[Cycle 1 Day 1]

Cmax AUClast

AUC24 tlast

[Cycle 1 Day 22]

Cmax tmax C24

AUC24 AUClast R(AUC24)

R(Cmax) CL/F tlast

Visit: Cycle 1 Day 1 and Cycle 1 Day 22 (Safety Evaluation Lead-in Part)

Analytical Method(s):

The following summaries will be provided for each analyte by visit.

(1) Descriptive statistics (mean, standard deviation, minimum, median and maximum) for PK parameters will be provided. In addition, geometric mean, 1<sup>st</sup> and 3<sup>rd</sup> quartiles, %CV, and geometric %CV will be computed for all PK parameters.

## 7.9.2 Pharmacodynamic Analysis

Not applicable

#### 7.10 **Other Outcomes**

Not applicable

#### 7.11 **Safety Analysis**

#### 7.11.1 **Adverse Events**

7.11.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

**Analysis** 

Variable(s): Treatment-emergent adverse event (TEAE)

[Related, Not Related] Categories: Relationship to Study Drug

Analytical

Method(s): The following summaries will be provided.

(1) Overview of Treatment-Emergent Adverse Events

- 1) All Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 2) Drug-related Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 3) Grade 3 or higher Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 4) Grade 3 or higher Drug-RelatedTreatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 5) Treatment-Emergent Adverse Events leading to study drug dose modification (number of events, number and percentage of subjects)
- Treatment-Emergent Adverse Events leading to study drug discontinuation (number of events, number and percentage of subjects)
- 7) Treatment-Emergent Adverse Events leading to study drug interruptions (number of events, number and percentage of subjects)
- Property of Takedai. For Treatment-Emergent Adverse Events leading to study drug reduction (number of events, number and percentage of subjects)

- 9) Serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 10) Drug-Related serious Treatment-Emergent Adverse Events (number of events, number and percentage of subjects)
- 11) Treatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)
- 12) Drug-RelatedTreatment-Emergent Adverse Events resulting in death (number of events, number and percentage of subjects)

TEAEs will be counted according to the rules below.

## Number of subjects

• Summaries for 2), 9), and 11)

A subject with occurrences of TEAE in both categories (ie, Related and Not Related) will be counted once in the Related category.

• Summary for 3) and 4)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum grade.

• Summaries other than 2), 3), 4), 9) and, 11)

A subject with multiple occurrences of TEAE will be counted only once.

## Number of events

For each summary, the total number of events will be calculated.

7.11.1.2 Frequency of patients with DLTs during Cycle 1 in the safety evaluation lead-in part.

Analysis Set: DLT population (For the refractory patients)

Analysis

Variable(s) Patients with DLTs during Cycle 1 [Yes, No]

Analytical

Method(s): Frequency distributions for categorical variables will be provided.

7.11.1.3 Displays of Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

## Categories:

Time of Onset (day)

[1 <= - <= 14, 15 <= - <= Max]ided using frequent (A and will)

Time of Onset for ILD/Pneumonitis Treatment-Emergent Adverse Events (day)

## Analytical Method(s):

The following summaries will be provided using frequency distribution.

TEAEs will be coded using the MedDRA and will be summarized using SOC and PT.

SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. SOC and PT will be sorted in decreasing frequency for tables provided by System Organ Class only or PT only.

- Treatment-Emergent Adverse Events by System Organ Class and (1) Preferred Term
- Treatment-Emergent Adverse Events by System Organ Class (2)
- Treatment-Emergent Adverse Events by Preferred Term (3)
- **(4)** Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Grade 3 or higher Treatment-Emergent Adverse Events by System (5) Organ Class and Preferred Term
- Grade 3 or higher Drug-Related Treatment-Emergent Adverse Events by System Organ Class, and Preferred Term
- Treatment-Emergent Adverse Events Leading to study drug modification by System Organ Class and Preferred Term
- Property of Takeda (8)Drug-Related Treatment-Emergent Adverse Events Leading to study drug modification by System Organ Class and Preferred Term
  - Treatment-Emergent Adverse Events leading to study drug dose (9) discontinuation by System Organ Class and Preferred Term
  - Drug-Related Treatment-Emergent Adverse Events Leading to (10)study drug discontinuation by System Organ Class and Preferred

- Class and Preferred Term

  I reatment-Emergent Adverse Events Leading to Term

  Treatment-Emergent Adverse Events Leading to System Organ Class and Preferred Term

  (13) Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term

  (14) Drug-Related Treatment-Emergent Adverse Events study drug reduction by System Organ Cristian System Organ Cristian System Organ Cristian Serious Treatment-Emergent Adverse Events Study drug reduction by System Organ Cristian S

- (16) Drug-Related Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (17) Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (18) Drug-Related Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (19) Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over Time
- (20) ILD/Pneumonitis Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (21) ILD/Pneumonitis Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Over Time
- (22) AED/Pneumonitis Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- ILD/Pneumonitis Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Property of Takeda. ILD/Pneumonitis Grade 3 or higher Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
  - (25) ILD/Pneumonitis serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
  - (26) ILD/Pneumonitis serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

- ILD/Pneumonitis Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (28) ILD/Pneumonitis Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- ILD/Pneumonitis Treatment-Emergent Adverse Events leading to (29)study drug discontinuation by System Organ Class and Preferred Term
- (30) ILD/Pneumonitis Treatment-Emergent Adverse Events leading to study drug interruptions by System Organ Class and Preferred Term
- (31) ILD/Pneumonitis Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term
- ILD/Pneumonitis Treatment-Emergent Adverse Events resulting (32)in death by System Organ Class and Preferred Term
- (33) ILD/Pneumonitis Drug-Related Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (34) Hypertension Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (35) Hypertension Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Hypertension Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Hypertension Drug-Related Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Hypertension serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (39)Hypertension serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (40) Hypertension Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Property of Takedai. (41) Hypertension Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

- Hypertension Treatment-Emergent Adverse Events leading to study drug discontinuation by System Organ Class and Preferred Term
- (43) Hypertension Treatment-Emergent Adverse Events leading to study drug interruptions by System Organ Class and Preferred Term
- (44) Hypertension Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term
- (45) Hypertension Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (46) Hypertension Drug-Related Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (47) Bradvcardia Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (48) Bradycardia Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (49) Bradycardia Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (50) Bradycardia Drug-Related Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (51) Bradycardia serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Bradycardia serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Bradycardia Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Property of Takedai. Bradycardia Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
  - Bradycardia Treatment-Emergent Adverse Events leading to study drug discontinuation by System Organ Class and Preferred Term
  - (56) Bradycardia Treatment-Emergent Adverse Events leading to study drug interruptions by System Organ Class and Preferred Term
  - (57)Bradycardia Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term
  - Bradycardia Treatment-Emergent Adverse Events resulting in

- death by System Organ Class and Preferred Term
- Bradycardia Drug-Related Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (60) GI Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (61) GI Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (62) GI Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (63) GI Drug-Related Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (64) GI serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (65) GI serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (66) GI Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (67) GI Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (68) GI Treatment-Emergent Adverse Events leading to study drug discontinuation by System Organ Class and Preferred Term
- GI Treatment-Emergent Adverse Events leading to study drug (69)interruptions by System Organ Class and Preferred Term
- GI Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term
- Property of Takedai. GI Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
  - GI Drug-Related Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
  - (73) Pancreatic Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
  - (74) Pancreatic Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
  - (75) Pancreatic Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

- (76)Pancreatic Drug-Related Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (77) Pancreatic serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (78) Pancreatic serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (79) Pancreatic Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (80) Pancreatic Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred
- (81) Pancreatic Treatment-Emergent Adverse Events leading to study drug discontinuation by System Organ Class and Preferred Term
- (82) Pancreatic Treatment-Emergent Adverse Events leading to study drug interruptions by System Organ Class and Preferred Term
- (83) Pancreatic Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term
- (84) Pancreatic Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (85) Pancreatic Drug-Related Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (86) Increased Insulin/Hyperglycemia Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (87) Increased Insulin/Hyperglycemia Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Property of Lakedai. (88) Increased Insulin/Hyperglycemia Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
  - Increased Insulin/Hyperglycemia Drug-Related Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
  - Increased Insulin/Hyperglycemia serious Treatment-Emergent (90)Adverse Events by System Organ Class and Preferred Term
  - (91) Increased Insulin/Hyperglycemia serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred

Term

- (92) Increased Insulin/Hyperglycemia Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (93) Increased Insulin/Hyperglycemia Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (94) Increased Insulin/Hyperglycemia Treatment-Emergent Adverse Events leading to study drug discontinuation by System Organ Class and Preferred Term
- (95) Increased Insulin/Hyperglycemia Treatment-Emergent Adverse Events leading to study drug interruptions by System Organ Class and Preferred Term
- (96) Increased Insulin/Hyperglycemia Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term
- (97) Increased Insulin/Hyperglycemia Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (98) Increased Insulin/Hyperglycemia Drug-Related Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (99) Hepatic Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (100) Hepatic Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (101) Hepatic Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (102) Hepatic Drug-Related Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (103) Hepatic serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (104) Hepatic serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (105) Hepatic Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

- (106) Hepatic Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (107) Hepatic Treatment-Emergent Adverse Events leading to study drug discontinuation by System Organ Class and Preferred Term
- (108) Hepatic Treatment-Emergent Adverse Events leading to study drug interruptions by System Organ Class and Preferred Term
- (109) Hepatic Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term
- (110) Hepatic Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (111) Hepatic Drug-Related Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (112) Elevated CPK Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (113) Elevated CPK Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (114) Elevated CPK Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (115) Elevated CPK Drug-Related Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (116) Elevated CPK serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (117) Elevated CPK serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (118) Elevated CPK Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Property of Lakeda. (119) Elevated CPK Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
  - (120) Elevated CPK Treatment-Emergent Adverse Events leading to study drug discontinuation by System Organ Class and Preferred
  - (121) Elevated CPK Treatment-Emergent Adverse Events leading to study drug interruptions by System Organ Class and Preferred

Term

- (122) Elevated CPK Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term
- (123) Elevated CPK Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (124) Elevated CPK Drug-Related Treatment-Emergent Adverse Events resulting in death by System Organ Class and Preferred Term
- (125) Visual Impairment Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (126) Visual Impairment Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (127) Visual Impairment Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (128) Visual Impairment Drug-Related Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (129) Visual Impairment serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (130) Visual Impairment serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (131) Visual Impairment Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (132) Visual Impairment Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Property of Lakedai. Visual Impairment Treatment-Emergent Adverse Events leading to study drug discontinuation by System Organ Class and Preferred Term
  - (134) Visual Impairment Treatment-Emergent Adverse Events leading to study drug interruptions by System Organ Class and Preferred Term
  - (135) Visual Impairment Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred
  - (136) Muscle Toxicity Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

- (137) Muscle Toxicity Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (138) Muscle Toxicity Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (139) Muscle Toxicity Drug-Related Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (140) Muscle Toxicity serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (141) Muscle Toxicity serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (142) Muscle Toxicity Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (143) Muscle Toxicity Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (144) Muscle Toxicity Treatment-Emergent Adverse Events leading to study drug discontinuation by System Organ Class and Preferred Term
- (145) Muscle Toxicity Treatment-Emergent Adverse Events leading to study drug interruptions by System Organ Class and Preferred Term
- (146) Muscle Toxicity Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term
- (147) Peripheral Neuropathy Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (148) Peripheral Neuropathy Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (149) Peripheral Neuropathy Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Property of Lakeda. (150) Peripheral Neuropathy Drug-Related Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
  - (151) Peripheral Neuropathy serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
  - (152) Peripheral Neuropathy serious Drug-Related Treatment-Emergent

- Adverse Events by System Organ Class and Preferred Term
- (153) Peripheral Neuropathy Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (154) Peripheral Neuropathy Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Preferred Term
- (155) Peripheral Neuropathy Treatment-Emergent Adverse Events leading to study drug discontinuation by System Organ Class and Preferred Term
- (156) Peripheral Neuropathy Treatment-Emergent Adverse Events leading to study drug interruptions by System Organ Class and Preferred Term
- (157) Peripheral Neuropathy Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term
- (158) Skin and Subcutaneous Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (159) Skin and Subcutaneous Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (160) Skin and Subcutaneous Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (161) Skin and Subcutaneous Drug-Related Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (162) Skin and Subcutaneous serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (163) Skin and Subcutaneous serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (164) Skin and Subcutaneous Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- Property of Takedai. (165) Skin and Subcutaneous Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
  - (166) Skin and Subcutaneous Treatment-Emergent Adverse Events leading to study drug discontinuation by System Organ Class and

#### Preferred Term

- (167) Skin and Subcutaneous Treatment-Emergent Adverse Events leading to study drug interruptions by System Organ Class and Preferred Term
- (168) Skin and Subcutaneous Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term
- (169) Photosensitivity Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (170) Photosensitivity Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (171) Photosensitivity Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (172) Photosensitivity Drug-Related Grade 3 or higher Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (173) Photosensitivity serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (174) Photosensitivity serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (175) Photosensitivity Grade 3 or higher serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (176) Photosensitivity Grade 3 or higher serious Drug-Related Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (177) Photosensitivity Treatment-Emergent Adverse Events leading to study drug discontinuation by System Organ Class and Preferred Term
- (178) Photosensitivity Treatment-Emergent Adverse Events leading to study drug interruptions by System Organ Class and Preferred Term
- (179) Photosensitivity Treatment-Emergent Adverse Events leading to study drug reduction by System Organ Class and Preferred Term
- Property of Lakedai. (180) Most commonly reported Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
  - (181) Most commonly reported Grade 3 or higher Treatment-Emergent

Adverse Events by System Organ Class and Preferred Term

(182) Most commonly reported Non-Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term

The frequency distribution will be provided according to the rules below.

## Number of subjects

analysis set.

Summary tables other than the CTCAE grade, (19), and (21) A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety

Summary tables for the CTCAE grade

A subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once for the TEAE with the maximum intensity. Percentages will be based on the number of subjects in the safety analysis set.

Summary table for (19) and (21)

A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC or a PT will be counted only once in that SOC or PT. When calculating percentages for each time interval, the number of subjects at risk (ie, subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.

Property of Takedai. Summary table for (180) and (181)

Most commonly reported TEAEs refer to PTs whose percentages are at least 10.0% in any one of the treatment groups.

Summary table for (182)

Most commonly reported Non-Serious TEAEs refer to PTs whose percentages are at least 5.0% in any one of the treatment groups. If no Non-Serious TEAEs exceed a frequency of 5.0%, the frequency cutoff of 2.0% will be used instead. Percentages will be based on the number of subjects in the safety analysis set.

# the applicable terms of Use 7.11.1.4 Time to Onset and the Duration of Special Interest Treatment-Emergent Adverse Events

Analysis Set: Safety Analysis Set

**Analysis** 

Variable(s): Time to initial onset of ILD/Pneumonitis

Time to initial onset of Bradycardia Even

Time to initial onset of Hypertension Eve

Time to initial onset of GI Events

Time to initial onset of Pancreatic Events

Time to initial onset of Increased Insulin/Hyperglycemia Events

Time to initial onset of Hepatic Events

Time to initial onset of Elevated CPK Events

Time to initial onset of Visual Impairment Events

Time to initial onset of Muscle Toxicity Events

Time to initial onset of Peripheral Neuropathy Events

Time to initial onset of Skin and Subcutaneous Events

Time to initial onset of Photosensitivity Events

Analytical

Method(s): For each variable, descriptive statistics will be provided.

#### Displays of Pretreatment Events 7.11.1.5

Analysis Set: All Subjects Who Signed the Informed Consent Form

**Analysis** 

Variable(s)

Pretreatment event (PTE)

Analytical

Method(s):

The following summaries will be provided using frequency distribution.

PTEs will be coded using the MedDRA and will be summarized using SOC and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency.

- (1) Pretreatment Events by System Organ Class and Preferred Term
- (2) Serious Pretreatment Events by System Organ Class and Preferred

Term

The frequency distribution will be provided according to the rules below.

## Number of subjects

s of the applicable since applicable is estable. A subject with multiple occurrences of PTE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of PTE within a PT will be counted only once in that PT.

#### 7.11.2 **Clinical Laboratory Evaluations**

#### 7.11.2.1 Hematology and Serum Chemistry

Analysis Set: Safety Analysis Set

**Analysis** 

Variable(s):

Hematology

Hematocrit

Platelet count Hemoglobin

White blood cell count with differential (ANC, basophils, eosinophils,

lymphocytes, monocytes)

**Serum Chemistry** 

Phosphorus

Alkaline phosphatase Albumin **Amylase** 

(ALP)

**ALT AST** Blood urea nitrogen

(BUN)

Calcium Bicarbonate (or total Creatine

> Phosphokinase (CPK) carbon dioxide)

Chloride Creatinine Glucose (fasted)

Lactate dehydrogenase C-reactive protein Magnesium

(LDH) (CRP)

> Potassium Sodium

Bilirubin (total bilirubin, conjugated and unconjugated bilirubin)

Protein (total protein) Uric acid HbA1c

Insulin Testosterone (Male Lipase

Patients Only)

Baseline, Cycle 1 Day 15, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6,

Cycle 7, Cycle 8, Cycle 9, Cycle 10, Cycle 11, Cycle 12, Cycle 13, Cycle 14, Cycle 15, Cycle 16, Cycle 17, Cycle 18 (except HbA1c and Testosterone)

Baseline, Cycle 4, Cycle 7, Cycle 10, Cycle 13, Cycle 16 (HbA1c)

Baseline, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6, Cycle 7, Cycle 8, Cycle 9, Cycle 10, Cycle 11, Cycle 12, Cycle 13, Cycle 14, Cycle 15, Cycle 16, Cycle 17, Cycle 18 (Testosterone)

## Analytical

Method(s):

For each variable, summaries (1) to (2) will be provided.

For applicable variables, summaries (3) will be provided.

(1) Summary of Laboratory Test Results and Change from Baseline by Visit

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

(2) Case Plots
Plots Over Time for each subject will be presented.

(3) Summary of Shifts of Laboratory Test Results
Shift tables will be generated showing changes in NCI CTCAE
grade from baseline to the worst postbaseline value.

## 7.11.3 Vital Signs

7.11.3.1 Vital Signs and Weight

Analysis Set: Safety Analysis Set

Analysis

Variable(s):

Systolic Blood Pressure

Diastolic Blood Pressure

Pulse

Respiratory rate

SpO2

Body temperature

Weight

Vicit.

Baseline, Cycle 1 Day8, Day 15, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6, Cycle 7, Cycle 8, Cycle 9, Cycle 10, Cycle 11, Cycle 12, Cycle 13, Cycle 14, Cycle 15, Cycle 16, Cycle 17, Cycle 18

Analytical

Method(s): For each variable, summaries (1) to (3) will be provided.

For applicable variables, summaries (4) will be provided.

(1) Summary of Vital Signs Parameters and Change from Baseline by Visit

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

(2) Case Plots

Plots over time for each subject will be presented.

(3) Summary of Shifts of Vital Signs Parameters
Shift tables will be generated showing changes in NCICTCAE grade from baseline to the worst postbaseline value.

### 7.11.4 12-Lead ECGs

Analysis Set: Safety Analysis Set

Analysis

Variable(s): 12-Lead ECG Interpretation [Within Normal Limits, Abnormal but not

Clinically Significant, Abnormal and

Clinically Significant]

**QT** Interval

**QTcF** Interval

Visit: Baseline, Cycle 2, Cycle 3, Cycle 4, Cycle 5, Cycle 6, Cycle 7, Cycle 8,

Cycle 9, Cycle 10, Cycle 11, Cycle 12, Cycle 13, Cycle 14, Cycle 15,

Cycle 16, Cycle 17, Cycle 18

Analytical

Method(s):

For each variable other than 12-lead ECG interpretations, summaries (1) and (2) will be provided.

For applicable variables, summary (3) will be provided.

For 12-lead ECG interpretation, summary (4) will be provided.

- (1) Summary of ECG Parameters and Change from Baseline by Visit Descriptive statistics for observed values and changes from baseline will be provided for each visit.
- (2) Case Plots
  Plots over time for each subject will be presented.
- (3) Number and Percentage of Subjects with Markedly Abnormal Values of ECG Parameters

to the applicable reims of Use Overall frequency distributions of MAV during treatment period will be provided. If an ECG laboratory parameter has both lower and upper MAV criteria, analysis will be performed for each. Further details are given in Appendix.

(4) Summary of Shift of 12-lead ECG Interpretation Shift table showing the number of subjects in each category at baseline and each post-baseline visit will be provided.

#### 7.11.5 **Other Observations Related to Safety**

Not applicable

#### 7.12 **Interim Analysis**

In this study, a 2-stage design will be used. An interim analysis for both futility and efficacy will be conducted in Stage 1, according to H1-minimax design in Englert. The proportion of patients achieving a confirmed objective response, per IRC, will be used as the endpoint for the interim analysis. The interim analysis will be performed with the first 29 patients in the main cohort of the expansion part at the cycle 6 after entry of the 29th patient. Enrollment will not be suspended during evaluation of these 29 patients; however, patients enrolled after the 29th patient in the main cohort of the expansion part will not be included in the interim analysis even if their ORR results were available on the cutoff date.

If the number of patients with confirmed ORR is 3 or fewer of the 29 patients, enrollment will be stopped entirely for futility. Additionally, if the number of patients with confirmed ORR is 10 or more of the 29 patients, it will be decided that brigatinib has demonstrated sufficient efficacy to reject the null hypothesis and declare superiority to the uninteresting ORR of 15% but the result at the timing of primary analysis will be interpreted descriptively. Otherwise, the study will continue until the 47 patients have had the opportunity to complete the Cycle 6 disease assessment. For the primary analysis, if the number of patients with confirmed ORR at the primary analysis is more than the number determined by the number at the interim analysis mentioned in Table 7.b, it will be decided that brigatinib has demonstrated sufficient efficacy to reject the null s. Ot sed. a. hypothesis. Of note, for the first 29 patients, their efficacy evaluation at the interim analysis were

Table 7.b Minimum Number of Confirmed ORR at the Primary Analysis

| No. ORR at Interim Analysis | No. ORR at Primary Analysis | |
|-----------------------------|-----------------------------|-------|
| 4/29 | 13/47 | all. |
| 5/29 | 13/47 | 70 |
| 6/29 | 13/47 | 0 |
| 7/29 | 13/47 | - 30° |
| 8/29 | 13/47 | dio |
| 9/29 | 12/47 | ~0K |

An IDMC will be formed. The IDMC will provide recommendation on the go/no go decision to move from the safety evaluation lead-in part to the expansion part, and on the futility and efficacy assessments performed at the interim analysis.

Furthermore for the publishment, the analysis only in safety lead-in part will be performed when all patients in safety lead-in part have had the opportunity to complet the cycle 6.

## 7.12.1 Analysis plan at the Interim Analysis

The analysis plan at interim analysis is based on this document except the following things.

- 1. The definition of FAS-P is a subset of the FAS population consisting of first 29 patients in the main cohort of the expansion part.
- 2. The point estimate mentioned in section 7.8.1.1 will be calculated based on the maximum likelihood estimation.
- 3. The interim analysis will be done for the all subjects who enroll the study until first 29 patients in the main cohort of the expansion part enroll the study.

## 7.12.2 Analysis plan in safety lead-in part

The analysis plan will be done as follows in 9 patients in safety lead-in part instead of analysis population specified in SAP.

- 1. Same analysis as section 7.4, 7.7, 7.8.1.2, 7.8.2.1, 7.9.1.2, 7.11.1.1, and 7.11.1.2 will be performed.
- 2. Same analysis as (1) and (3) in section 7.9.1.1 will be performed.
- 3. Same analysis as (1), (4), (5), (6), (9), (10), (11), (12), (13), (14), (15), (16), and (17) in section 7.11.1.3 will be performed.
- 4. The analysis for best response in target lesions in section 7.8.2.3 will be performed.

Tianned Analysis for the Refractory Patients

The analysis for the refractory patients will be performed when all refractory patients have had the opportunity to complete the Cycle 7 Day 1 disease assessment. The data for TKI-naïve Patients will be excluded from the analysis.

7.13.2 Planned 4--1

The analysis for TKI-naïve Patients will be performed after the final database lock at the end of the study. For efficacy and pharmacokinetic analysis, the same analysis described in section 7.8 to 7.9 as the one for the refractory patients will be performed only in TKI-naïve Patient. Additionally, 12 months PFS rate as assessed by an IRC, per RECIST version 1.1 in the TKInaïve expansion cohort will be performed as primary endpoint. For disposition of subjects, demographic, compliance, and safety analysis, the same analysis described in section 7.3 to 7.7, and 7.11 as the one for the refractory patients will be performed in TKI-naïve Patient and in all patients who have been enrolled.

#### 7.13.3 **Planned Final Analysis**

For efficacy analysis, the analysis described in section 7.8 to 7.9 will be performed in following population.

- TKI-naïve Patients.
- Refractory Patients.

For disposition of subjects, demographic, compliance, and safety analysis, the same analysis described in section 7.3 to 7.7, and 7.11 will be performed in following population

- TKI-naïve Patients.
- Refractory Patients
- All patients who have been enrolled.

#### 7.14 **Changes in the Statistical Analysis Plan**

Based on comment from the team members, the following things has been changed.

- The analysis for photosensitivity event as special interest AE has been added.
- The analysis which was done in adhoc analysis has been added as additional analysis.
- Section 7.13.3 has been added.

EORTC QLQ-C30 Scoring Manual (3rd edition). Fayers PM Acre
Groenvold M, Curran D, Bottomley A. on bok-10
EORTC, 2001. ISBN: 2,0200

shimoz .ational Inst. Ikeda S, Shiroiwa T, Igarashi A, Noto S, Fukuda T, and Saito S, Shimozuma K. Developing a Japanese version of the EQ-5D-5L value set. Journal of the National Institute of Public Health,

## Appendix 1 Criteria for Markedly Abnormal Values

For each parameter except upper MAV Criteria of QTcF Interval, all evaluable data (ie, non-missing data) will be classified as a MAV or not. The criteria in the table below will be used.

For each parameter and subject, classifications will be made according to the conditions i) to in provided below. The lower and the upper criteria will be considered separately.

- i) A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- ii) A subject who does not meet condition i) and has at least one evaluable data after baseline that doesn't meet the MAV criteria will be considered as a subject without MAV.
- iii) A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV for that parameter.

#### 12-lead ECG

| | MAV | MAV Criteria |
|----------------------|----------------|----------------|
| Parameter | Lower Criteria | Upper Criteria |
| QT Interval (msec) | <=50 | >=460 |
| QTcF Interval (msec) | <=50 | - |

For upper MAV Criteria of QTcF Interval, all evaluable data (ie, non-missing data) will be classified as a MAV or not. The criteria in the table below will be used. Note that the observed value and the change from baseline used for classification should be measurements taken on the same day.

For each subject, classifications will be made according to the conditions i) to iii) provided below.

- i) A subject with at least one evaluable data after baseline that meets the MAV criteria will be classified as a subject with MAV.
- ii) A subject who does not meet condition i) and has at least one evaluable data after baseline that meets any of the following will be considered as a subject without MAV.
  - Observed value is less than 450 msec and not missing.
  - Change from baseline is less than 30 msec and not missing, and observed value is less than 500 msec and not missing.
- iii) A subject who does not meet conditions i) or ii) will be excluded from the analysis of MAV.

| | | MAV Criteria |
|---|---|---|
| Parameter | Lower Criteria | Upper Criteria |
| QTcF Interval (msec) - | | If either of the following conditions is met: |
| | | • observed value >=500 |
| | | • change from baseline >= 30 and observed value |
| Stakeda. For n | on recommercial. | If either of the following conditions is met: • observed value >= 500 • change from baseline >= 30 and observed value ≥ change from baseline >= 30 and observed value ≥ description of the following conditions is met: • observed value >= 500 • change from baseline >= 30 and observed value ≥ description of the following conditions is met: • observed value >= 500 • change from baseline >= 30 and observed value ≥ description of the following conditions is met: • observed value >= 500 • change from baseline >= 30 and observed value ≥ description of the following conditions is met: • observed value >= 500 • change from baseline >= 30 and observed value ≥ description of the following conditions is met: • observed value >= 500 • change from baseline >= 30 and observed value ≥ description of the following conditions is met: • observed value >= 500 • change from baseline >= 30 and observed value ≥ description of the following conditions is met: • observed value >= 500 description of the following conditions is met: description of the f |

# Appendix 2 Definition of Adverse Event of GI events, Hepatic events and Visual Impairment Events

• GI events

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| SMQ: Gastrointestinal | 10000059 | Abdominal discomfort |
| nonspecific symptoms and | 10000060 | Abdominal distension |
| therapeutic procedures — | 10000081 | Abdominal pain |
| _ | 10000084 | Abdominal pain lower |
| _ | 10000087 | Abdominal pain upper |
| | 10060926 | Abdominal symptom |
| | 10000097 | Abdominal tenderness |
| _ | 10063541 | Bowel movement irregularity |
| _ | 10008399 | Change of bowel habit |
| _ | 10010774 | Constipation |
| | 10012735 | Diarrhoea |
| | 10079120 | Discoloured vomit |
| _ | 10053155 | Epigastric discomfort |
| | 10015137 | Eructation |
| | 10016766 | Flatulence |
| | 10017367 | Frequent bowel movements |
| | 10017999 | Gastrointestinal pain |
| | 10067715 | Gastrointestinal sounds abnormal |
| | 10059024 | Gastrointestinal toxicity |
| 77 | 10059158 | Infrequent bowel movements |
| For hour Coll | 10028813 | Nausea |
| ~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~ | 10062501 | Non-cardiac chest pain |
| _ | 10053634 | Oesophageal discomfort |
| _ | 10030180 | Oesophageal pain |
| _ | 10047700 | Vomiting |
| Other PTs | 10013950 | Dysphagia |
| _ | 10070840 | Gastrointestinal tract irritation |
| Other PTs | 10067171 | Regurgitation |
| | 10038776 | Retching |
| | 10047708 | Vomiting projectile |

(a) MedDRA version 23.0.

## Hepatic events

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| SMQ: Liver related<br>investigations, signs and<br>symptoms | 10001547 | Alanine aminotransferase abnormal |
| | 10001551 | Alanine aminotransferase increased |
| | 10003477 | Aspartate aminotransferase abnormal |
| | 10003481 | Aspartate aminotransferase increased |
| | 10067718 | Bilirubin conjugated abnormal |
| | 10004685 | Bilirubin conjugated increased |
| | 10077356 | Bilirubin urine present |
| | 10004792 | Biopsy liver abnormal |
| | 10058477 | Blood bilirubin abnormal |
| | 10005364 | Blood bilirubin increased |
| | 10005370 | Blood bilirubin unconjugated increased |
| | 10078360 | Computerised tomogram liver abnorma |
| | 10052554 | Foetor hepaticus |
| _ | 10059710 | Galactose elimination capacity test abnormal |
| | 10059712 | Galactose elimination capacity test decreased |
| | 10017688 | Gamma-glutamyltransferase abnormal |
| | 10017693 | Gamma-glutamyltransferase increased |
| _ | . 10051333 | Guanase increased |
| | 10019621 | Hepaplastin abnormal |
| | 10019622 | Hepaplastin decreased |
| | 10068997 | Hepatic artery flow decreased |
| COT | 10062685 | Hepatic enzyme abnormal |
| | 10060794 | Hepatic enzyme decreased |
| , O' — | 10060795 | Hepatic enzyme increased |
| | 10019670 | Hepatic function abnormal |
| | 10067365 | Hepatic hydrothorax |
| <i>√</i> 0. | 10076254 | Hepatic hypertrophy |
| | 10057110 | Hepatic mass |
| X 21- | 10019705 | Hepatic pain |
| _ | 10066244 | Hepatic sequestration |
| <u></u> | 10068358 | Hepatic vascular resistance increased |
| Kakedai. For non-com | 10066195 | Hepatobiliary scan abnormal |
| | 10019842 | Hepatomegaly |
| _ | 10019847 | Hepatosplenomegaly |
| | 10020575 | Hyperammonaemia |
| | 10020578 | Hyperbilirubinaemia |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| | 10051924 | Hypercholia |
| | 10068237 | Hypertransaminasaemia |
| | 10024690 | Liver function test abnormal |
| | 10077677 | Liver function test decreased |
| | 10077692 | Liver function test increased |
| | 10052550 | Liver induration |
| | 10075895 | Liver palpable |
| | 10061947 | Liver scan abnormal |
| | 10024712 | Liver tenderness |
| | 10064712 | Mitochondrial aspartate aminotransferas increased |
| | 10049631 | Oedema due to hepatic disease |
| | 10054125 | Perihepatic discomfort |
| | 10067338 | Retrograde portal vein flow |
| | 10064558 | Total bile acids increased |
| | 10062688 | Transaminases abnormal |
| | 10054889 | Transaminases increased |
| | 10045428 | Ultrasound liver abnormal |
| | 10050792 | Urine bilirubin increased |
| | 10056536 | X-ray hepatobiliary abnormal |
| | 10059571 | Blood alkaline phosphatase abnormal |
| | 10059570 | Blood alkaline phosphatase increased |
| | 10071634 | Deficiency of bile secretion |
| | 10049483 | Glutamate dehydrogenase increased |
| <u> </u> | 10080824 | Glycocholic acid increased |
| , , , O | 10059766 | Haemorrhagic ascites |
| ,0 | 10074084 | Hepatic fibrosis marker abnormal |
| No. | 10074413 | Hepatic fibrosis marker increased |
| <b>K</b> 0 | 10079686 | Hepatic lymphocytic infiltration |
| 70. | 10020942 | Hypoalbuminaemia |
| EQ. | 10077291 | Model for end stage liver disease score abnormal |
| keda. For hones | 10077292 | Model for end stage liver disease score increased |
| | 10068821 | Periportal oedema |
| | 10069000 | Peritoneal fluid protein abnormal |
| | 10068999 | Peritoneal fluid protein decreased |
| | 10068998 | Peritoneal fluid protein increased |
| | 10082832 | AST/ALT ratio abnormal |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| | 10084058 | Congestive hepatopathy |
| _ | 10083172 | Hepatic venous pressure gradient abnormal |
| _ | 10083171 | Hepatic venous pressure gradient increased |
| _ | 10084071 | Liver opacity |
| _ | 10083123 | Magnetic resonance imaging liver abnormal |
| SMQ: Cholestasis and jaundice | 10061009 | Bilirubin excretion disorder |
| of hepatic origin | 10048611 | Cholaemia |
| _ | 10008635 | Cholestasis |
| _ | 10067969 | Cholestatic liver injury |
| _ | 10064190 | Cholestatic pruritus |
| _ | 10072268 | Drug-induced liver injury |
| _ | 10019754 | Hepatitis cholestatic |
| _ | 10020578 | Hyperbilirubinaemia |
| _ | 10021209 | Icterus index increased |
| _ | 10023126 | Jaundice |
| | 10023129 | Jaundice cholestatic |
| _ | 10023136 | Jaundice hepatocellular |
| | 10066758 | Mixed liver injury |
| _ | 10058117 | Ocular icterus |
| | 10074151 | Parenteral nutrition associated liver disease |
| _ | 10071634 | Deficiency of bile secretion |
| | 10048245 | Yellow skin |
| SMQ: Hepatic failure, fibrosis | 10080860 | Acquired hepatocerebral degeneration |
| and cirrhosis and other liver | 10000804 | Acute hepatic failure |
| damage-related conditions | 10077305 | Acute on chronic liver failure |
| | 10070815 | Acute yellow liver atrophy |
| <i>√</i> 0, − | 10003445 | Ascites |
| _ | 10003547 | Asterixis |
| _ | 10068547 | Bacterascites |
| <i>~</i> . − | 10004659 | Biliary cirrhosis |
| _ | 10004664 | Biliary fibrosis |
| 7 OK | 10082480 | Cardiohepatic syndrome |
| _ | 10067969 | Cholestatic liver injury |
| _ | 10057573 | Chronic hepatic failure |
| damage-related conditions | 10010075 | Coma hepatic |
| _ | 10063075 | Cryptogenic cirrhosis |
| _ | 10071265 | Diabetic hepatopathy |
| _ | 10072268 | Drug-induced liver injury |
| | 10051010 | Duodenal varices |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|-------------------|-------------|------------------------------------|
| | 10072319 | Gallbladder varices |
| - | 10076237 | Gastric variceal injection |
| - | 10076238 | Gastric variceal ligation |
| - | 10051012 | Gastric varices |
| - | 10057572 | Gastric varices haemorrhage |
| _ | 10061997 | Hepatectomy |
| _ | 10019637 | Hepatic atrophy |
| - | 10065274 | Hepatic calcification |
| - | 10019641 | Hepatic cirrhosis |
| - | 10019660 | Hepatic encephalopathy |
| _ | 10066599 | Hepatic encephalopathy prophylaxis |
| - | 10019663 | Hepatic failure |
| - | 10019668 | Hepatic fibrosis |
| - | 10067365 | Hepatic hydrothorax |
| - | 10064668 | Hepatic infiltration eosinophilic |
| - | 10061998 | Hepatic lesion |
| - | 10019692 | Hepatic necrosis |
| - | 10077215 | Hepatic steato-fibrosis |
| _ | 10019708 | Hepatic steatosis |
| - | 10019772 | Hepatitis fulminant |
| _ | 10062000 | Hepatobiliary disease |
| _ | 10053244 | Hepatocellular foamy cell syndrome |
| - | 10019837 | Hepatocellular injury |
| - | 10052274 | Hepatopulmonary syndrome |
| CO. | 10019845 | Hepatorenal failure |
| - C/10 - | 10019846 | Hepatorenal syndrome |
| ,0, - | 10019851 | Hepatotoxicity |
| - 0(, ) | 10071502 | Intestinal varices |
| - | 10078058 | Intestinal varices haemorrhage |
| 70. | 10076640 | Liver dialysis |
| - | 10024670 | Liver disorder |
| - | 10067125 | Liver injury |
| - | 10062040 | Liver operation |
| - | 10024714 | Liver transplant |
| kedai. For non-co | 10025129 | Lupoid hepatic cirrhosis |
| - | 10076204 | Minimal hepatic encephalopathy |
| - | 10066758 | Mixed liver injury |
| - | 10051081 | Nodular regenerative hyperplasia |
| - | 10082249 | Nonalcoholic fatty liver disease |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| | 10053219 | Non-alcoholic steatohepatitis |
| | 10077259 | Non-cirrhotic portal hypertension |
| | 10049631 | Oedema due to hepatic disease |
| | 10030210 | Oesophageal varices haemorrhage |
| | 10073215 | Peripancreatic varices |
| | 10074726 | Portal fibrosis |
| | 10036200 | Portal hypertension |
| | 10079446 | Portal hypertensive colopathy |
| | 10068923 | Portal hypertensive enteropathy |
| | 10050897 | Portal hypertensive gastropathy |
| | 10073979 | Portal vein cavernous transformation |
| | 10073209 | Portal vein dilatation |
| | 10067281 | Portopulmonary hypertension |
| | 10080429 | Primary biliary cholangitis |
| | 10080679 | Regenerative siderotic hepatic nodule |
| | 10052279 | Renal and liver transplant |
| | 10067338 | Retrograde portal vein flow |
| | 10039012 | Reye's syndrome |
| | 10070953 | Reynold's syndrome |
| | 10067823 | Splenic varices |
| | 10068662 | Splenic varices haemorrhage |
| | 10076331 | Steatohepatitis |
| | 10056956 | Subacute hepatic failure |
| <u></u> | 10056091 | Varices oesophageal |
| CO. | 10072284 | Varicose veins of abdominal wall |
| | 10078438 | White nipple sign |
| ~O. — | 10083521 | Immune-mediated hepatic disorder |
| MQ: Hepatitis, non-infectious | 10066263 | Acute graft versus host disease in liver |
| | 10071198 | Allergic hepatitis |
| <i>─</i> | 10080576 | Alloimmune hepatitis |
| | 10003827 | Autoimmune hepatitis |
| - X 3/C | 10072160 | Chronic graft versus host disease in live |
| _ | 10008909 | Chronic hepatitis |
| MQ: Hepatitis, non-infectious | 10064676 | Graft versus host disease in liver |
| | 10019717 | Hepatitis |
| _ | 10019727 | Hepatitis acute |
| | 10019754 | Hepatitis cholestatic |
| | 10019755 | Hepatitis chronic active |
| | 10019759 | Hepatitis chronic persistent |

| PT_CODE (a) | PT_NAME (a) |
|---|---|
| 10019772 | Hepatitis fulminant |
| 10019795 | Hepatitis toxic |
| 10078962 | Immune-mediated hepatitis |
| 10023025 | Ischaemic hepatitis |
| 10067737 | Lupus hepatitis |
| 10053219 | Non-alcoholic steatohepatitis |
| 10051015 | Radiation hepatitis |
| 10076331 | Steatohepatitis |
| | 10019772<br>10019795<br>10078962<br>10023025<br>10067737<br>10053219<br>10051015 |

(a) MedDRA version 23.0.

## • Visual Impairment Events

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| HLGT: vision disorder | 10000389 | Accommodation disorder |
| - | 10001902 | Amaurosis |
| - | 10001903 | Amaurosis fugax |
| - | 10001906 | Amblyopia |
| - | 10001912 | Amblyopia strabismic |
| - | 1000191 | Amblyopia tobacco |
| - | 10002534 | Aniseikonia |
| - | 10002537 | Anisometropia |
| - | 10003569 | Astigmatism |
| - | 10005169 | Blindness |
| - | 10005177 | Blindness cortical |
| 3 | 10005178 | Blindness day |
| CO | 10005184 | Blindness transient |
| 000 | 10005186 | Blindness unilateral |
| . 100 | 10008585 | Chloropsia |
| \\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | 10008795 | Chromatopsia |
| - | 10010051 | Colour blindness acquired |
| 9,0 | 10012646 | Diabetic blindness |
| - | 10013036 | Diplopia |
| <b>∠</b> ⊘′ − | 10013892 | Dyschromatopsia |
| ·<br>· | 10015290 | Erythropsia |
| Takedai. For non-con- | 10019099 | Halo vision |
| - | 10020675 | Hypermetropia |
| - | 10028651 | Myopia |
| - | 10029404 | Night blindness |
| - | 10034962 | Photopsia |
| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| | 10036628 | Presbyopia |
| | 10038264 | Refraction disorder |
| | 10038266 | Refractive amblyopia |
| | 10039677 | Scintillating scotoma |
| | 10042441 | Sudden visual loss |
| | 10044245 | Toxic optic neuropathy |
| | 10047511 | Vision abnormal neonatal |
| | 10047513 | Vision blurred |
| | 10047531 | Visual acuity reduced |
| | 10047532 | Visual actify reduced transiently |
| | 10047571 | Visual impairment |
| | 10048216 | Xanthopsia |
| | 10049155 | Visual brightness |
| | 10051819 | Cyanopsia |
| | 10052087 | Oscillopsia |
| | 10052128 | Glare |
| | 10053549 | Altered visual depth perception |
| | 10059397 | Antimetropia |
| | 10061322 | Optic nerve disorder |
| | 10061323 | Optic neuropathy |
| | . 10063341 | Metamorphopsia |
| | 10063354 | Charles Bonnet syndrome |
| | 10064133 | Loss of visual contrast sensitivity |
| | 10067557 | Dysmetropsia |
| C | 10068906 | Computer vision syndrome |
| | 10070917 | Eccentric fixation |
| 100 | 10072729 | Delayed dark adaptation |
| 1.0 | 10073286 | Pathologic myopia |
| akedai. For non-cs | 10074928 | Low luminance best-corrected visual acuit decreased |
| 100 | 10075919 | Pseudomyopia |
| Sie | 10076241 | Psychogenic visual disorder |
| | 10076302 | Optic nerve compression |
| | 10076660 | Cortical visual impairment |
| | 10078300 | Acute myopia |
| | 10078508 | Homonymous diplopia |
| | 10078509 | Heteronymous diplopia |
| | 10079450 | Visual snow syndrome |
| | 10079805 | Delayed light adaptation |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| | 10081186 | Central vision loss |
| SMQ: retinal disorder | 10054881 | Acquired pigmented retinopathy |
| _ | 10079367 | Acute macular outer retinopathy |
| | 10074444 | Acute zonal occult outer retinopathy |
| | 10064930 | Age-related macular degeneration |
| _ | 10001903 | Amaurosis fugax |
| | 10002444 | Angiogram retina abnormal |
| _ | 10063452 | Arteriosclerotic retinopathy |
| _ | 10071578 | Autoimmune retinopathy |
| _ | 10004390 | Benign neoplasm of retina |
| _ | 10072959 | Birdshot chorioretinopathy |
| _ | 10008762 | Chorioretinal atrophy |
| <del>-</del> | 10061763 | Chorioretinal disorder |
| _ | 10008766 | Chorioretinal scar |
| _ | 10008769 | Chorioretinitis |
| _ | 10063118 | Chorioretinopathy |
| _ | 10010050 | Colour blindness |
| _ | 10010051 | Colour blindness acquired |
| <del>-</del> | 10010056 | Colour vision tests abnormal |
| _ | 10010057 | Colour vision tests abnormal blue-yellow |
| _ | 10010058 | Colour vision tests abnormal red-green |
| _ | 10071321 | Commotio retinae |
| _ | 10058202 | Cystoid macular oedema |
| -2 | 10079805 | Delayed light adaptation |
| Takedai. For non-cod | 10071004 | Detachment of macular retinal pigment epithelium |
| , O' — | 10052501 | Detachment of retinal pigment epithelium |
| _ | 10012688 | Diabetic retinal oedema |
| _ | 10012689 | Diabetic retinopathy |
| | 10078228 | Diffuse uveal melanocytic proliferation |
| _ | 10075567 | Dry age-related macular degeneration |
| - A 21/2 | 10015831 | Extraocular retinoblastoma |
| _ | 10015901 | Exudative retinopathy |
| | 10051045 | Eye naevus |
| _ | 10017520 | Fundoscopy abnormal |
| _ | 10081899 | Hypotony maculopathy |
| _ | 10077392 | Immune recovery uveitis |
| _ | 10073499 | Internal limiting membrane peeling |
| _ | 10073929 | IRVAN syndrome |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| | 10059239 | Leukaemic retinopathy |
| | 10049935 | Lipaemia retinalis |
| | 10025407 | Macular cyst |
| | 10025409 | Macular degeneration |
| | 10075873 | Macular detachment |
| | 10071392 | Macular fibrosis |
| | 10051058 | Macular hole |
| | 10065534 | Macular ischaemia |
| | 10025415 | Macular oedema |
| | 10025416 | Macular opacity |
| | 10071041 | Macular pigmentation |
| | 10060815 | Macular pseudohole |
| | 10025419 | Macular reflex abnormal |
| | 10065319 | Macular rupture |
| | 10063185 | Macular scar |
| | 10081199 | Macular telangiectasia |
| | 10025425 | Maculopathy |
| | 10026432 | Malignant neoplasm of retina |
| | 10063341 | Metamorphopsia |
| | 10079959 | Myopic chorioretinal degeneration |
| | 10080534 | Myopic traction maculopathy |
| | 10064997 | Necrotising retinitis |
| | 10071129 | Neovascular age-related macular degeneration |
| Fornonia | 10062940 | Neuropathy, ataxia, retinitis pigmentosa syndrome |
| 2011 | 10074696 | Noninfective chorioretinitis |
| | 10074699 | Noninfective retinitis |
| ₹o. | 10081568 | Non-proliferative retinopathy |
| vý. | 10065311 | Paraneoplastic retinopathy |
| COC | 10034962 | Photopsia |
| , at | 10037525 | Pupillary light reflex tests abnormal |
| | 10075189 | Purtscher retinopathy |
| (akedai. Foil) | 10064714 | Radiation retinopathy |
| | 10064145 | Retinal aneurysm |
| | 10079121 | Retinal aneurysm rupture |
| | 10038824 | Retinal arteriovenous malformation |
| | 10038826 | Retinal artery embolism |
| | 10038827 | Retinal artery occlusion |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|--------------------|-------------|---------------------------------|
| | 10038829 | Retinal artery spasm |
| | 10038830 | Retinal artery stenosis |
| | 10038831 | Retinal artery thrombosis |
| | 10077911 | Retinal collateral vessels |
| | 10052643 | Retinal coloboma |
| | 10074908 | Retinal cryoablation |
| | 10038839 | Retinal cyst |
| | 10038840 | Retinal cyst excision |
| | 10038845 | Retinal degeneration |
| | 10038846 | Retinal depigmentation |
| | 10038847 | Retinal deposits |
| | 10038848 | Retinal detachment |
| | 10038853 | Retinal disorder |
| | 10062776 | Retinal drusen |
| | 10038857 | Retinal dystrophy |
| | 10038862 | Retinal exudates |
| | 10071391 | Retinal fibrosis |
| | 10038866 | Retinal function test abnormal |
| | 10038867 | Retinal haemorrhage |
| | 10067848 | Retinal implant |
| | . 0051742 | Retinal infarction |
| | 10064833 | Retinal infiltrates |
| | 10057430 | Retinal injury |
| | 10038871 | Retinal ischaemia |
| C | 10038873 | Retinal laser coagulation |
| | 10057428 | Retinal melanocytoma |
| 70. | 10038878 | Retinal melanoma |
| | 10052784 | Retinal migraine |
| | 10057407 | Retinal neoplasm |
| <b>%</b> 0. | 10055666 | Retinal neovascularisation |
| To. | 10038886 | Retinal oedema |
| | 10062107 | Retinal operation |
| | 10038891 | Retinal pallor |
| akedai. For non-co | 10071246 | Retinal perivascular sheathing |
| | 10069652 | Retinal phototoxicity |
| | 10062971 | Retinal pigment epithelial tear |
| | 10038893 | Retinal pigment epitheliopathy |
| | 10038894 | Retinal pigmentation |
| | 10038895 | Retinal scar |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|-----------------|-------------|--------------------------------------|
| | 10038897 | Retinal tear |
| | 10038899 | Retinal telangiectasia |
| | 10077890 | Retinal thickening |
| | 10048955 | Retinal toxicity |
| | 10067870 | Retinal transplant |
| | 10038900 | Retinal tumour excision |
| | 10038901 | Retinal vascular disorder |
| | 10038903 | Retinal vascular occlusion |
| | 10062108 | Retinal vascular thrombosis |
| | 10038905 | Retinal vasculitis |
| | 10038907 | Refinal vein occlusion |
| | 10038908 | Retinal vein thrombosis |
| | 10081463 | Retinal vein varices |
| | 10073562 | Retinal vessel avulsion |
| | 10079569 | Retinal white without pressure |
| | 10038910 | Retinitis |
| | 10038914 | Retinitis pigmentosa |
| | 10038916 | Retinoblastoma |
| | 10059663 | Retinogram abnormal |
| | 10038923 | Retinopathy |
| | 10051447 | Retinopathy haemorrhagic |
| | 10038926 | Retinopathy hypertensive |
| | 10038930 | Retinopathy hyperviscosity |
| | 10038933 | Retinopathy of prematurity |
| S | 10038934 | Retinopathy proliferative |
| | 10038935 | Retinopathy sickle cell |
| ,00 | 10038936 | Retinopathy solar |
| Fot bourge | 10066985 | Retinopexy |
| | 10061492 | Retinoschisis |
| 80. | 10065569 | Rhegmatogenous retinal detachment |
| LO | 10039677 | Scintillating scotoma |
| < 01 | 10066785 | Scleral buckling surgery |
| Kakeda: For | 10040114 | Serous retinal detachment |
| | 10081652 | Serpiginous choroiditis |
| | 10062958 | Subretinal fibrosis |
| | 10069356 | Subretinal fluid |
| | 10071935 | Subretinal haematoma |
| | 10082240 | Subretinal hyperreflective exudation |
| | 10080316 | Tractional retinal detachment |

| Search criteria | PT CODE (a) | DT NAME (a) |
|---|---|---|
| Search Criteria | = 17 | PT_NAME (a) Tunnel vision |
| | 10045178 | |
| | 10065622 | Venous stasis retinopathy Visual field tests abnormal |
| | 10047567 | |
| | 10066421 | Vitreal cells |
| | 10047644 | Vitrectomy |
| | 10071035 | Vitreomacular interface abnormal |
| | 10057435 | Vitreous adhesions |
| | 10047650 | Vitreous detachment |
| | 10047651 | Vitreous disorder |
| | 10047654 | Vitreous floaters |
| | 10071936 | Vitreous haematoma |
| | 10047655 | Vitreous haemorrhage |
| | 10077514 | Vitreous haze |
| | 10047663 | Vitritis |
| | 10081123 | Autoimmune eye disorder |
| | 10005169 | Blindness |
| | 10005184 | Blindness transient |
| | 10005186 | Blindness unilateral |
| | 10081186 | Central vision loss |
| | 10008795 | Chromatopsia |
| | 10081428 | Ciliary body melanoma |
| | 10013892 | Dyschromatopsia |
| | 10015916 | Eye disorder |
| | 10079891 | Eye haematoma |
| C | 10015926 | Eye haemorrhage |
| | 10078394 | Eye opacity |
| 10 | 10081445 | Foveal reflex abnormal |
| 1.0 | 10077000 | Hypertensive cerebrovascular disease |
| | 10071934 | Intraocular haematoma |
| 70. | 10081061 | Intra-ocular injection complication |
| TO. | 10076430 | Intravitreal implant |
| ( Die | 10053150 | Leukocoria |
| (akedai. For non.co | 10074928 | Low luminance best-corrected visual acuit decreased |
| | 10069385 | Ocular ischaemic syndrome |
| | 10075324 | Ocular lymphoma |
| | 10082039 | Ocular stem cell transplant |
| | 10081144 | Ophthalmic artery thrombosis |
| | 10074349 | Ophthalmic vein thrombosis |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| | 10073561 | Optical coherence tomography abnormal |
| · | 10034051 | Pars plana cyst |
| - | 10073286 | Pathologic myopia |
| - | 10034960 | Photophobia |
| · | 10074603 | Red reflex abnormal |
| - | 10081068 | Sclerotomy |
| - | 10071573 | Susac's syndrome |
| - | 10081431 | Uveal melanoma |
| - | 10047513 | Vision blurred |
| - | 10047531 | Visual acuity reduced |
| • | 10047534 | Visual acuity tests abnormal |
| - | 10047555 | Visual field defect |
| • | 10047571 | Visual impairment |
| - | 10082001 | Vogt-Koyanagi-Harada disease |
| - | 10048216 | Xanthopsia |
| | 10071989 | Vascular endothelial growth factor overexpression |
| • | 10082802 | Disruption of the photoreceptor inner segment-outer segment |
| - | 10083006 | Eye infarction |
| - | 10083087 | Fluorescence angiogram abnormal |
| - | 10083329 | Foveal degeneration |
| - | 10082768 | Hyperaesthesia eye |
| - | 10083069 | Immune-mediated uveitis |
| · · | 10082596 | Optic disc traction syndrome |
| ,00 | 10083565 | Orbital haematoma |
| 0// | 10083187 | Serous retinopathy |
| - | 10083502 | Tessellated fundus |
| Forhonico | 10083563 | Transpupillary thermotherapy |
| 1 steps. Fo | 10031045 | Orbital haemorrhage |
| 9.00 | 10048896 | Retinal fovea disorder |
| · X | 10071181 | Vitreoretinal traction syndrome |
| | 10001902 | Amaurosis |
| SMQ: glaucoma | 10001903 | Amaurosis fugax |
| • | 10071364 | Anterior chamber angle neovascularisation |
| • | 10069166 | Blebitis |
| • | 10005169 | Blindness |
| - | | |
| | 10005178 | Blindness day |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| | 10005186 | Blindness unilateral |
| | 10007739 | Cataract |
| • | 10061769 | Ciliary body operation |
| | 10069165 | Conjunctival filtering bleb leak |
| | 10080692 | Coreoplasty |
| | 10079171 | Deep anterior chamber of the eye |
| | 10072729 | Delayed dark adaptation |
| • | 10014456 | Electrooculogram abnormal |
| • | 10074027 | Exfoliation syndrome |
| | 10072289 | Eye colour change |
| | 10057105 | Eye laser surgery |
| | 10015958 | Eye pain |
| , | 10016059 | Facial pain |
| | 10052128 | Glare |
| , | 10077986 | Goniotomy |
| | 10022943 | Iridoschisis |
| , | 10022948 | Iris atrophy |
| | 10057420 | Iris operation |
| | 10074928 | Low luminance best-corrected visual acuit decreased |
| | 10068960 | Narrow anterior chamber angle |
| | 10029404 | Night blindness |
| | 10030041 | Ocular hyperaemia |
| | <u> </u> | Ophthalmic artery thrombosis |
| -0 | 10074349 | Ophthalmic vein thrombosis |
| 2,0 | 10048544 | Ophthalmodynamometry abnormal |
| 2011 | 10061321 | Optic disc disorder |
| | 10034546 | Periorbital pain |
| ₹O, | 10034960 | Photophobia |
| \\ \dots\\\ \dots\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\\ | 10037520 | Pupillary block |
| .00 | 10059663 | Retinogram abnormal |
| 1 Stores | 10081068 | Sclerotomy |
| stakedai. For non-co | 10067126 | Seidel test positive |
| )' | 10066418 | Tenon's cyst |
| | 10047513 | Vision blurred |
| | 10047531 | Visual acuity reduced |
| | 10047532 | Visual acuity reduced transiently |
| | 10047549 | Visual evoked potentials abnormal |
| | 10047571 | Visual impairment |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| | 10082768 | Hyperaesthesia eye |
| | 10083516 | Iris discolouration |
| SMQ: lens disorder | 10054045 | Anterior capsule contraction |
| _ | 10063937 | Capsular block syndrome |
| | 10008795 | Chromatopsia |
| _ | 10012369 | Deposit eye |
| | 10078228 | Diffuse uveal melanocytic proliferation |
| _ | 10013892 | Dyschromatopsia |
| _ | 10078394 | Eye opacity |
| _ | 10024203 | Lens dislocation |
| _ | 10061219 | Lens disorder |
| _ | 10071370 | Lens extraction |
| _ | 10052980 | Lenticular operation |
| _ | 10074928 | Low luminance best-corrected visual acui decreased |
| | 10082039 | Ocular stem cell transplant |
| _ | 10074603 | Red reflex abnormal |
| | 10047513 | Vision blurred |
| _ | 10047531 | Visual acuity reduced |
| | 10047571 | Visual impairment |
| other PTs | 10000173 | Abnormal sensation in eye |
| | 10071684 | Anterior chamber collapse |
| _ | 10002683 | Anterior chamber opacity |
| ~ | 10070497 | Aqueous humour leakage |
| co <del>,</del> | 10003552 | Asthenopia |
| | 10081123 | Autoimmune eye disorder |
| ·20, — | 10008422 | Chemical burns of eye |
| _ | 10010804 | Contact lens intolerance |
| _ | 10012369 | Deposit eye |
| ~~· | 10013774 | Dry eye |
| _ | 10015911 | Eye burns |
| - 2k | 10015916 | Eye disorder |
| _ | 10015943 | Eye inflammation |
| Takedai. For non-co | 10061128 | Eye injury |
| | 10015946 | Eye irritation |
| | 10078394 | Eye opacity |
| <del>-</del> | 10081699 | Eye pH abnormal |
| <del>-</del> | 10081700 | Eye pH decreased |
| | 10081701 | Eye pH increased |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|----------------------|-------------|---------------------------------------|
| | 10073423 | Eye ulcer |
| | 10016760 | Flat anterior chamber of eye |
| | 10051116 | Foreign body sensation in eyes |
| | 10074563 | Graft versus host disease in eye |
| | 10020939 | Hypoaesthesia eye |
| | 10072139 | Ocular rosacea |
| | 10082449 | Ocular surface squamous neoplasia |
| | 10061137 | Ocular toxicity |
| | 10056836 | Ophthalmological examination abnormal |
| | 10034960 | Photophobia |
| | 10042530 | Superficial injury of eye |
| | 10073692 | Fear break up time decreased |
| | 10049267 | Thermal burns of eye |
| | 10061412 | Vitamin A deficiency eye disorder |
| | 10048221 | Xerophthalmia |
| | 10001903 | Amaurosis fugax |
| | 10001906 | Amblyopia |
| | 10003230 | Arteritis |
| | 10075688 | Autoimmune demyelinating disease |
| | 10081123 | Autoimmune eye disorder |
| | . 010005169 | Blindness |
| | 10005184 | Blindness transient |
| | 10005185 | Blindness traumatic |
| | 10005186 | Blindness unilateral |
| G | 10081186 | Central vision loss |
| | 10008087 | Cerebral arteritis |
| 70. | 10008795 | Chromatopsia |
| | 10010051 | Colour blindness acquired |
| . < | 10010056 | Colour vision tests abnormal |
| 70. | 10061094 | Cranial nerve injury |
| TE . | 10072729 | Delayed dark adaptation |
| X OL | 10076456 | Delayed myelination |
| | 10012305 | Demyelination |
| Kakedai. For hon. co | 10013892 | Dyschromatopsia |
| | 10049020 | Encephalitis periaxialis diffusa |
| | 10015923 | Eye excision |
| | 10061852 | Eye operation |
| | 10069060 | Eye prosthesis insertion |
| | 10069061 | Eye prosthesis removal |

| Search criteria | PT_CODE (a) | PT_NAME (a) |
|---|---|---|
| | 10017520 | Fundoscopy abnormal |
| | 10019452 | Hemianopia |
| • | 10019455 | Hemianopia heteronymous |
| | 10019456 | Hemianopia homonymous |
| | 10077000 | Hypertensive cerebrovascular disease |
| • | 10064133 | Loss of visual contrast sensitivity |
| • | 10074928 | Low luminance best-corrected visual acu decreased |
| | 10029404 | Night blindness |
| | 10069385 | Ocular ischaemic syndrome |
| | 10081144 | Ophthalmic artery thrombosis |
| | 10056836 | Ophthalmological examination abnorma |
| • | 10030949 | Optic pathway injury |
| | 10065372 | Orbitotomy |
| | 10077820 | Quadrantanopia |
| • | 10063613 | Radiotherapy to eye |
| | 10038956 | Retro-orbital neoplasm |
| | 10039677 | Scintillating scotoma |
| | 10045178 | Tunnel vision |
| | 10067485 | Uhthoff's phenomenon |
| | 10047531 | Visual acuity reduced |
| • | 10047532 | Visual acuity reduced transiently |
| | 10047534 | Visual acuity tests abnormal |
| | 10047555 | Visual field defect |
| c.O | 10047567 | Visual field tests abnormal |
| , <u>, , </u> | 10047571 | Visual impairment |
| (a) MedDRA version 23.0. | 10061411 | Visual pathway disorder |
| | 10061412 | Vitamin A deficiency eye disorder |

## Photosensitivity

| E (a) | PT_NAME (a | PT_CODE (a) | Search criteria |
|---|---|---|---|
| urigo | Actinic prurig | 10000616 | ll PTs of HLT: Photosensitivity |
| sease | Hartnup diseas | 10019165 | and photodermatosis conditions |
| geruption | Juvenile spring eru | 10023269 | |
| y reaction | Photosensitivity re | 10034972 | |
| ht eruption | Polymorphic light e | 10036087 | |
| natitis | Solar dermatit | 10041303 | |
| n | Sunburn | 10042496 | |
| atosis | Photodermatos | 10051246 | |
| nsitivity reaction | Injection site photosensiti | 10053396 | _ |
| ensitivity reaction | Application site photosensi | 10058730 | _ |
| nsitivity reaction | Infusion site photosensiti | 10065486 | _ |
| stosis | Actinic elastos | 10068388 | _ |
| dermatitis | Chronic actinic der | 10072578 | |
| osensitivity | Implant site photoser | 10073415 | |
| | Administration site photosen | 10075961 | |
| | Medical device site photosen | 10076137 | |
| <u> </u> | Vaccination site photosensi | 10076186 | |
| • | Hydroa vaccinifo | 10083442 | |
| | | | Takeda. For non-com |
| | | | Lakega. |

## ELECTRONIC SIGNATURES

| ELECTRONIC SIGNATURES | | |
|---|---|---|
| Signed by | Meaning of Signature | Server Date (dd-MMM-yyyy HH, mm 'UTC') |
| PPD | | (dd-MM-yyyy H-H-min CTC) |
| Signed by PPD Signed by PPD PPD Signed by PPD PPD Signed by PPD | ercial use only and subject | io ine appri |